## CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

DMID Protocol: 13-0053 Study Title:

A Phase I, Single Dose, Open-label, Study Comparing the Pharmacokinetics and Safety of Pretomanid in Subjects with Mild, Moderate, and Severe Hepatic Impairment to Matched, Non-Hepatically Impaired Subjects

NCT02422524

Version 2.0

**DATE: 08 May 2024** 

RESTRICTED

## STUDY TITLE

| Protocol Number Code: | DMID Protocol: 13-0053 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | Pretomanid |
| Form/Route: | Tablet/Oral |
| Indication Studied: | Tuberculosis |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | First subject enrolled 29MAR2018 (screened 19MAR) |
| Clinical Trial Completion Date: | |
| Date of the Analysis Plan: | 08 May 2024 |
| Version Number: | 2.0 |

## This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# **VERSION HISTORY**

| SAP Version | Change | Rationale |
|---|---|---|
| 1.0 | Not Applicable | Original version. |
| 2.0 | Removed "sequential" when describing the order of group enrollments based on changes to the study design (i.e., simultaneous enrollment allowed in the moderate and severe groups). | The study protocol was amended after finalization of<br>the SAP v1.0. These SAP updates were driven by<br>protocol changes, including the addition of a second<br>site (Saint Louis). |
| | "PA-824" replaced with "Pretomanid" throughout to align with the protocol. | |
| | Added language to clarify the definition of baseline in Section 6.1: "In general, the last recorded value prior to study drug administration will be considered as baseline." | |
| | Section 6.2 was updated to adjust the planned timing of interim analyses to align with protocol v7.0. | |
| | Updated Section 6.7, Section 10.3, added additional tables, and expanded others to account for by-site summaries and analyses following the addition of the Saint Louis site. | |
| | Updated eligibility criteria listed throughout to align with protocol v7.0. | |
| | Updated Table 3: Schedule of Study Procedures and Figure 2: Schematic of Study Design to align with protocol v7.0. | |
| | Updated Table 5: Laboratory/Clinical Adverse Event Grading Scale to align with the protocol v7.0. | |

# TABLE OF CONTENTS

| STUDY | TITLE | II |
|---|---|---|
| VERSIC | ON HISTORY | III |
| TABLE | OF CONTENTS | IV |
| LIST O | F ABBREVIATIONS | VII |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 2.1. | Purpose of the Analyses | 2 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. | Study Objectives | 3 |
| 3.1.1. | Primary Study Objective | 3 |
| 3.1.2. | Primary Study Objective | 3 |
| 3.2. | Endpoints | 3 |
| 3.2.1. | Primary Outcome Measures | 3 |
| 3.2.2. | Secondary Outcome Measures | 3 |
| 3.3. | Study Definitions and Derived Variables | 4 |
| 3.3.1. | Impairment Group Definitions | 4 |
| 4. | INVESTIGATIONAL PLAN | 5 |
| 4.1. | Overall Study Design and Plan | 5 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 5 |
| 4.3. | Selection of Study Population | 5 |
| 4.3.1. | Study Inclusion Criteria | 5 |
| Inclusion | n Criteria for Patients with Hepatic Impairment (Groups 1-3) | 5 |
| Inclusion | n Criteria for Non-Hepatically Impaired Controls (Group 4) | 6 |
| 4.3.2. | Study Exclusion Criteria | 7 |
| Exclusion | on Criteria for Patients with Hepatic Impairment (Groups 1-3) | 7 |
| Exclusion | on Criteria for Non-Hepatically Impaired Controls (Group 4) | 8 |
| 4.4. | Treatments | 10 |
| 4.4.1. | Treatments Administered | 10 |
| 4.4.2. | Identity of Investigational Product(s) | 10 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 10 |

#### **Table of Contents** (continued) 4.4.4. 4.4.5. 4.4.6. 4.4.7. 4.4.8. 4.5. 4.5.1. 4.5.2. Safety Variables 12 5. 6. 6.1. 6.2. Timing of Analyses 14 6.3. 6.3.1. 6.3.2. 6.4. 6.5. 6.6. Multicenter Studies 15 6.7. 6.8. 7. 7.1. Disposition of Subjects 16 7.2. Protocol Deviations \_\_\_\_\_\_\_16 8. 9. 9.1. Prior and Concurrent Medical Conditions 18 9.1.1. 9.1.2. 9.2. Measurements of Treatment Compliance 18 9.3. 9.3.1.

#### **Table of Contents** (continued) 9.4. 9.5. Pregnancies 19 9.6. 9.7. 9.8. 9.9. 10. 10.1. 10.2. 10.2.1. Concentration Summaries. 22 10.2.2. Pharmacokinetic Parameters 22 10.3. Comparison of Impairment Groups 23 11. 12. OTHER ANALYSES \_\_\_\_\_\_\_26 13. 14. TECHNICAL DETAILS......28 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED 16. REFERENCES 30 17. APPENDIX 1. TABLE MOCK-UPS.......35

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|---|---|
| ALT | Alanine Aminotransferase |
| ANOVA | Analysis of Variance |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Category |
| AUC | Area Under the Concentration-Time Curve |
| AUC <sub>(0-last)</sub> | AUC to the Last Measurable Concentration |
| $\mathrm{AUC}_{(0-\infty)}$ | AUC Extrapolated to Infinity |
| BUN | Blood Urea Nitrogen |
| С | Celsius |
| CBC | Complete Blood Count |
| CL/F | Apparent Oral Clearance |
| $C_{max}$ | Maximum Concentration |
| CI | Confidence Interval |
| CNS | Central Nervous System |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| CV | Coefficients of Variation |
| DHHS | Department of Health and Human Services |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| F | Fahrenheit |
| FDA | Food and Drug Administration |
| GM | Geometric Mean |
| HEENT | Head, Eyes, Ears, Nose and Throat |
| HDPE | High-density polyethylene |
| HBsAg | Hepatitis B surface antigen |
| HIV | Human Immunodeficiency Virus |

# **List of Abbreviations** (continued)

| ICH | International Conference on Harmonisation |
|---|---|
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ITT | Intention to Treat |
| $\lambda_z$ | Elimination Rate Constant |
| LLOQ | Lower Limit of Quantitation |
| max | maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| min | Minimum |
| mITT | Modified Intention to Treat |
| MRI | Magnetic Resonance Imaging |
| N | Number (typically refers to subjects) |
| NCA | Noncompartmental Analysis |
| NIAID | National Institute of Allergy and Infectious Diseases, NIH, DHHS |
| NIH | National Institutes of Health |
| OTC | Over the Counter |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PP | Per Protocol |
| PR | P-R Interval on an ECG |
| PT | Preferred Term |
| QT/QTc | QT Interval of an ECG/Corrected QT Interval of an ECG |
| QTcF | Heart Rate-Corrected QT Interval (Fridericia's Formula) |
| | R-squared Adjusted |
| $R_{adjusted}^2$ | |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| t <sub>(1/2)</sub> | Apparent Terminal Elimination Half-Life |

# **List of Abbreviations** (continued)

| $T_{\text{max}}$ | Time to Obtain Maximum Concentration (C <sub>max</sub> ) |
|-------------------|----------------------------------------------------------|
| ТВ | Tuberculosis |
| V <sub>d</sub> /F | Apparent Volume of Distribution During Terminal Phase |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "DMID Protocol 13-0053: A Phase 1, Single Dose, Open-label, Study Comparing the Pharmacokinetics and Safety of Pretomanid in Subjects with Mild, Moderate, and Severe Hepatic Impairment to Matched, Non-hepatically Impaired Subjects" describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses as well as all planned sample tables, listings and figures. Regarding the final analysis and final integrated Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines (1), as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials).

Any deviation from this statistical plan will be described and justified in the final study report, as appropriate. The reader of this SAP is encouraged to also review the clinical protocol for details on conduct of the study and the operational aspects of clinical assessments.

Some minor modifications may be necessary to the planned design of tables, figures, and listings to accommodate data collected during the actual study conduct.

## 2. INTRODUCTION

Tuberculosis (TB) causes a significant global health burden with an estimated annual worldwide incidence in 2015 of approximately 10.4 million new cases (2). Approximately 1.8 million people died from TB in 2015 (2, 3) making TB the leading infectious killer of adults worldwide. TB is also the leading infectious cause of death among people with HIV or acquired immunodeficiency syndrome (4).

TB is an infectious disease caused by the bacterium *Mycobacterium tuberculosis* (MTB). This infection primarily affects the lungs (pulmonary TB) but can affect other organs such as the kidneys, bones, and brain (5). TB is transmitted by inhalation of infective droplets containing MTB and expelled into the air by a person with active TB (5).

The mainstays of therapy against TB are antibiotic combination regimens. The recommended treatment includes a combination of rifampin, isoniazid, pyrazinamide, ethambutol or streptomycin (6 - 8). A 4-drug regimen of directly observed therapy is administered for 2 months (intensive phase) and is then followed by rifampin and isoniazid for an additional 4-7 months (7). The goal of the prolonged regimen is to ensure sterilization of tuberculosis lesions and to prevent development of drug resistance (8). If administered correctly, cure rates as high as 95% can be achieved (9).

Unfortunately, the prolonged and complicated treatment course of TB affects patient compliance (10), which has led to development of multi-drug resistant TB (MDR-TB) (7, 10) and extensively drug resistant strains (XDR-TB) (11). The WHO estimates that ~4% of new TB cases, and 20% of previously treated cases of TB have MDR-TB (4). Of those new MDR-TB cases 9% are XDR-TB (4). Therefore, there is a need to develop novel drugs, such as Pretomanid (previously known as PA-824) to be used in combination, for the treatment of TB.

In previous efficacy studies Pretomanid was shown to have bactericidal activity in a much shorter treatment time than the current recommended regimen. Table 2 shows a summary of previous phase 2 studies involving Pretomanid.

# 2.1. Purpose of the Analyses

Pretomanid is metabolized extensively in the liver (CYP3A4) and has a low extraction ratio. In the setting of advanced liver disease both hepatic blood flow and hepatic function can be compromised. Therefore, the pharmacokinetics of Pretomanid are likely to be altered in subjects with hepatic impairment compared to matched healthy subjects. The purpose of this protocol is to evaluate the safety and pharmacokinetics of Pretomanid in the setting of underlying liver disease defined as a Child-Pugh score of A, B, or C.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

## 3.1.1. Primary Study Objective

• To evaluate the pharmacokinetics of a single oral dose of Pretomanid in subjects with mild, moderate, and severe hepatic impairment (as assessed by Child-Pugh score), relative to matched non-hepatically impaired subjects.

#### 3.1.2. Primary Study Objective

 To evaluate the safety of a single oral dose of Pretomanid in subjects with mild, moderate, and severe hepatic impairment (as assessed by Child-Pugh score), relative to matched non-hepatically impaired subjects.

## 3.2. Endpoints

#### 3.2.1. Primary Outcome Measures

- The pharmacokinetics of a single-dose of Pretomanid will be assessed from serial blood samples collected prior to dosing (Day 1) and at multiple time points post dosing: 1 h, 2 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h, and 96 h. The primary outcome measure will be total plasma concentration of Pretomanid. The following will be determined:
  - $AUC_{(0-\infty)}$ : Area under the concentration time-curve extrapolated to infinity
  - AUC<sub>(0-last)</sub>: Area under the concentration time-curve to the last concentration above the lower limit of quantitation (LLOQ)
  - C<sub>max</sub>: Maximum Pretomanid concentration
  - T<sub>max</sub>: Time of maximum Pretomanid concentration
  - $t_{(1/2)}$ : Apparent terminal elimination half-life
  - CL/F: Apparent oral clearance calculated from Dose/AUC<sub>(0-∞)</sub>
  - V<sub>d</sub>/F: Apparent Volume of Distribution

## 3.2.2. Secondary Outcome Measures

- The secondary outcome measures will be:
  - Incidence and severity of serious adverse events reported at any time from the time of study treatment through the end of the study.
  - Incidence and severity of related adverse events at any time from the time of study treatment through Day 12.
  - Summary of physical examination findings (height at baseline, and weight at serial time points from Day of Admission until Day 12), vital signs (serial time points from Day of Admission

until Day 12), safety laboratory parameters (Day of Admission, as well as Days 2, 5, and 12), and ECG data (Day of Admission and Day 12).

## 3.3. Study Definitions and Derived Variables

Maximum plasma concentration ( $C_{max}$ ) is defined as: the maximum observed drug concentration in blood plasma for a particular dose interval.

Time of maximum plasma concentration ( $T_{max}$ ) is defined as: the time at which the maximum plasma concentration occurs.

Elimination rate constant ( $\lambda_z$ ) is defined as the first-order rate constant describing rate of elimination from plasma.

The apparent terminal elimination half-life (t(1/2)) will be estimated by ln(2) divided by  $\lambda_z$ .

AUC(0-last) is defined as the area under the concentration-time curve (AUC) from administration (time 0) to the time of the last quantifiable concentration above the LLOQ.

AUC(0- $\infty$ ) is defined as the total AUC and will be computed by adding AUC<sub>0-t</sub> to an extrapolated value equal to the last measured concentration greater than limits of quantitation divided by  $\lambda_z$  and will be calculated using

$$AUC_{0-\infty} = AUC_{0-t} + \frac{C_{tf}}{\lambda_Z},$$

where  $C_{tf}$  is the last measurable concentration  $\geq LLOQ$ 

Apparent oral clearance (CL/F) will be calculated as the dose divided by the AUC( $0-\infty$ ).

Apparent volume of distribution  $(V_d/F)$  is defined as: the theoretical volume that the total amount of administered drug would occupy to provide the same concentration as it currently is in blood plasma divided by the bioavailability.

$$V_d / F = \frac{Dose}{\lambda z \times AUC_{0-\infty}}$$

## 3.3.1. Impairment Group Definitions

Subjects are stratified into 4 groups based on the Child-Pugh score. The Child-Pugh score is based on five clinical measures of liver function: total bilirubin, serum albumin, prothrombin, ascites and hepatic encephalopathy. Based on their score (as determined by the site) patients are defined as mild hepatic impairment (5-6 points), moderate hepatic impairment (7-9 points), or severe hepatic impairment (10-15 points). The impairment group designations are:

- Mild Hepatic Impairment: Child-Pugh A (5-6 points)
- Moderate Hepatic Impairment: Child-Pugh B (7-9 points)
- Severe Hepatic Impairment: Child-Pugh C (10-15 points)
- Matched Controls: Non-hepatically impaired controls

## 4. INVESTIGATIONAL PLAN

## 4.1. Overall Study Design and Plan

Approximately 6 subjects will be enrolled in each of the hepatic impairment groups (Mild, Moderate and Severe), and approximately 18 non-hepatically impaired subjects will be enrolled as matched controls.

Subjects with hepatic impairment from all three groups will be enrolled starting with subjects who have mild hepatic impairment. Subjects with moderate and severe hepatic disease will be enrolled simultaneously. If enrollment into the severe hepatic impairment group is completed before that of the moderate hepatic impairment group, results from the severe cohort will be analyzed to determine the impact of severe hepatic impairment on the PK of Pretomanid and the need to continue enrollment of persons with moderate hepatic impairment will be reevaluated to determine whether the objectives of the study have been met. Non-hepatically impaired subject matches will be dosed only after the corresponding subject with hepatic impairment has completed the 36-hour blood sampling procedure. The group of up to 18 matched controls will be matched to the 18 subjects with hepatic impairment based on age ( $\pm$  10 years) and body weight at screening ( $\pm$  20% body weight). A control subject may be matched to more than one hepatic impairment subject if warranted, and if the subjects to which they are matched are not in the same disease severity group. Control subjects may be matched to hepatically impaired subjects at any site. Therefore, there may be less than 18 subjects with normal hepatic function (Table 1; Figure 2).

Subjects will receive a single oral dose of Pretomanid 200 mg taken with 240 mL of water after overnight fast.

## 4.2. Discussion of Study Design, Including the Choice of Control Groups

This is a Phase 1, single dose (200 mg), open-label, study comparing the pharmacokinetics and safety of Pretomanid in subjects with mild, moderate, and severe hepatic impairment relative to matched non-hepatically impaired subjects.

Non-hepatically impaired controls will be identified from the site specific registries and the community. Subjects for this study may also be identified through advertisement, letters, and other forms of communication.

# 4.3. Selection of Study Population

The study population will be representative of subjects with varying degrees of liver disease as defined by Child-Pugh scores. The Child-Pugh scores used for eligibility in the study will be calculated by the site at screening only.

#### 4.3.1. Study Inclusion Criteria

## **Inclusion Criteria for Patients with Hepatic Impairment (Groups 1-3)**

- 1. Subject is able to give voluntary written informed consent before any study related procedure is performed.
- 2. 18-70 years of age, inclusive.

- 3. Acceptable laboratory values\* obtained at screening (within 21 days prior to admission to the confinement/hospital unit) and at admission to the confinement/hospital unit.
  - \*Chemistry, complete blood count, AST, ALT, total bilirubin, alkaline phosphatase, albumin, and urinalysis deemed not clinically significant by the investigator.
- 4. Hepatic impairment classified as Child-Pugh class A (mild), B (moderate), or C (severe) criteria at screening for Groups 1, 2, or 3, respectively, and documented evidence of hepatic cirrhosis\*.
  - \*by biopsy, nuclear scan, CT, MRI, ultrasound, or other clinically acceptable methods
- 5. If female, not of childbearing potential\* or agrees to avoid becoming pregnant by using acceptable contraception\*\* during the duration of the study.
  - \*Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral oophorectomy or status after hysterectomy.
  - \*\*Females of childbearing potential must agree to use two acceptable methods of contraceptives: bilateral tubal ligation; barrier method (condom) by the male partner (even if vasectomized); hormonal contraceptives; intrauterine contraceptive devices; diaphragm in combination with contraceptive jelly, cream, foam, or spermicide; and abstinence from sexual intercourse with men.
- 6. If subject is male and capable of reproduction, agrees to avoid fathering a child for three months after dosing by using an acceptable method of birth control\*.
  - \*In addition to the use of a barrier method (condom) even if vasectomized, acceptable methods of birth control are restricted to a monogamous relationship with a woman who agrees to use acceptable contraception as outlined in inclusion criterion #5, and abstinence from sexual intercourse with women.
- 7. If the subject is female, a negative serum pregnancy test at screening and a negative urine pregnancy test at admission to confinement/hospital unit.
- 8. Willingness to comply with all protocol requirements.

## **Inclusion Criteria for Non-Hepatically Impaired Controls (Group 4)**

- 1. Subject is able to give voluntary written informed consent before any study related procedure is performed.
- 2. 18-70 years of age, inclusive.
- 3. Subject is a healthy volunteer as determined by no clinically significant findings from medical history, physical examination, vital signs, and 12-lead ECG as determined by the Site Investigator.
- 4. Acceptable laboratory values\* obtained at screening (within 21 days prior to admission to the confinement/hospital unit) and either at or within 72 hours of admission to the confinement/hospital unit.
  - \*Chemistry, complete blood count, AST, ALT, total bilirubin, alkaline phosphatase, albumin, and urinalysis within the reference range for the test laboratory, unless deemed not clinically significant by the investigator.
- 5. If female, not of childbearing potential\* or agrees to avoid becoming pregnant by using acceptable contraception\*\* during the duration of the study.
  - \*Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral oophorectomy or status after hysterectomy.
  - \*\*Females of childbearing potential must agree to use two acceptable methods of contraceptives: bilateral tubal ligation; barrier method (condom) by the male partner (even if vasectomized); hormonal contraceptives; intrauterine contraceptive

devices; diaphragm in combination with contraceptive jelly, cream, foam, or spermicide; and abstinence from sexual intercourse with men.

- 6. If subject is male and capable of reproduction, agrees to avoid fathering a child for three months after dosing by using an acceptable method of birth control\*.
  - \*In addition to the use of a barrier method (condom) even if vasectomized, acceptable methods of birth control are restricted to a monogamous relationship with a woman who agrees to use acceptable contraception as outlined in inclusion criterion #5, and abstinence from sexual intercourse with women.
- 7. If the subject is female, a negative serum pregnancy test at screening and a negative urine pregnancy test at admission to confinement/hospital unit.
- 8. Willingness to comply with all protocol requirements.

## 4.3.2. Study Exclusion Criteria

## **Exclusion Criteria for Patients with Hepatic Impairment (Groups 1-3)**

- 1. Hypokalemia (< 3.5mEq/L), severe hypomagnesemia (< 1.1 mg/dL) or severe hypocalcemia (< 7.5 mg/dL).
- 2. AST or ALT > 10 times the upper limit of normal.
- 3. Creatinine clearance < 60 ml/min.
- 4. Inability to swallow tablets.
- 5. Presence of any condition or finding\* which would jeopardize subject safety, impact study result validity, or diminish the subject's ability to undergo all study procedures and assessments\*\*.
  - \*in the opinion of the site investigator \*\*e.g., inability to draw PK samples
- 6. History of fever or documented fever (oral temperature  $\geq$ 100.4° F or  $\geq$  38.0° C) in the 48 hours prior to admission to the confinement/hospital unit.
- 7. Currently breastfeeding.
- 8. History of chronic tobacco/nicotine use (>10 cigarettes per day for 3 months minimum prior to confinement/hospital unit admission).
- 9. History of clinically significant allergy or severe side effects with nitroimidazoles (e.g., Metronidazole and related substances and azole antifungals or aromatase inhibitors).
- 10. Receipt of an investigational drug, vaccine or biologic in a clinical trial within 30 days prior to screening.
- 11. Use of any over the counter (OTC) medication\* within 7 days prior to admission to the confinement/hospital unit, unless\*\* the substance would not likely impact the validity of the study results.

<sup>\*</sup>including vitamins and herbal supplements, cough and cold medications.

<sup>\*\*</sup>in the opinion of the site investigator

12. Treatment with CYP450 enzyme altering drugs\* within 7 days prior to admission to the confinement/hospital unit, unless\*\* the substance would not likely impact the validity of the study results.

\*except hormonal contraceptives

\*\*in the opinion of the site investigator

NOTE: See list of CYP450 enzyme altering drugs under the concomitant medications Section 4.4.7.

- 13. A positive blood screen for HIV.
- 14. A positive alcohol breath test (or other suitable test for alcohol) or a urine screen test for drugs of abuse\* at screening and at admission to the confinement/hospital unit.

\*Amphetamines, barbiturates, cocaine metabolites, marijuana, opiates, phencyclidine (PCP).

NOTE: Results of the urine screen test can be ignored if in the opinion of the PI the results can be explained by the concomitant medications history.

- 15. Unwillingness to abstain from engaging in strenuous physical activity (e.g. running, bicycling, weightlifting, competitive sports) during the course of the study.
- 16. Consumption of grapefruit juice in the 48 hours before admission to the confinement/hospital unit, or the inability to abstain from these until completion of Day 12.
- 17. A QTcF interval >450 msec (males) or >450 msec (females) at screening (Visit 00A) or admission to the confinement/hospital unit (Visit 00B) or a history of prolonged QTc interval.
- 18. A family history\* of Long QT Syndrome, premature cardiac death\*\*, or sudden death without a preceding diagnosis of a condition\*\*\* that could be causative of sudden death.

\*parents

- \*\*due to ischemic heart disease or sudden cardiac death before 55 years of age (men) or 65 years of age (women)
- \*\*\*such as known coronary artery disease, congestive heart failure, or terminal cancer
- 19. Any clinically significant ECG abnormality, in the opinion of the site investigator, at screening and at admission to the confinement/hospital unit.
- 20. Donation of >500 mL blood within the 30 days prior to admission to the confinement/hospital unit.
- 21. Plans to donate blood during the study or up to 14 days after dosing.
- 22. Persons with a transjugular intrahepatic portosystemic shunt.

## **Exclusion Criteria for Non-Hepatically Impaired Controls (Group 4)**

- 1. Inability to swallow tablets.
- 2. Presence of any condition or finding\* which would jeopardize subject safety, impact study result validity, or diminish the subject's ability to undergo all study procedures and assessments\*\*.
  - \*in the opinion of the site investigator \*\*e.g., inability to collect PK samples
- 3. History of fever or documented fever (oral temperature  $\geq$ 100.4° F or  $\geq$  38.0° C) in the 48 hours prior to admission to the confinement/hospital unit.

- 4. Currently breastfeeding.
- 5. History of chronic tobacco/nicotine use (>10 cigarettes per day for 3 months minimum prior to confinement/hospital unit admission).
- 6. History of seizures (other than febrile seizures during childhood) or known or suspected CNS disorders that may predispose to seizures.
- 7. History of clinically significant allergy or severe side effects with nitroimidazoles (e.g., Metronidazole and related substances and azole antifungals or aromatase inhibitors).
- 8. Receipt of an investigational drug, vaccine or biologic in a clinical trial within 30 days prior to screening.
- 9. Use of any over the counter (OTC) medication\* within 7 days prior to admission to the confinement/hospital unit, unless\*\* the substance would not likely impact the validity of the study results.
  - \*including vitamins and herbal supplements, antacids, cough and cold medications.
  - \*\*in the opinion of the site investigator
- 10. Use of prescription medication except hormonal contraceptives within 30 days prior to admission to the confinement/hospital unit, unless\* the substance would not likely impact study result validity.
  - \*in the opinion of the site investigator
- 11. Treatment with CYP450 enzyme altering drugs\* within 7 days prior to admission to the confinement/hospital unit, unless\*\* the substance would not likely impact the validity of the study results.
  - \*except hormonal contraceptives
  - \*\*in the opinion of the site investigator

NOTE: See list of CYP450 enzyme altering drugs under the concomitant medications Section 4.4.7.

- 12. A positive blood screen for HIV.
- 13. A positive blood screen for hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
- 14. A positive alcohol breath test (or other suitable test for alcohol) or a urine screen test for drugs of abuse\* at screening and at admission to the confinement/hospital unit.
  - \*Amphetamines, barbiturates, benzodiazepines, cocaine metabolites, marijuana, opiates, phencyclidine (PCP).
- 15. A history of alcohol abuse or dependence within the past 1 month prior to admission to the confinement/hospital unit.
- 16. Unwillingness to abstain from engaging in strenuous physical activity (e.g. running, bicycling, weightlifting, competitive sports) during the course of the study.
- 17. Consumption of grapefruit juice in the 48 hours before admission to the confinement/hospital unit, or the inability to abstain from these until completion of Day 12.

- 18. A QTcF interval >450 msec (males) or >450 msec (females) at screening (Visit 00A) or admission to the confinement/hospital unit (Visit 00B) or a history of prolonged QTc interval.
- 19. A family history\* of Long QT Syndrome, premature cardiac death\*\*, or sudden death without a preceding diagnosis of a condition\*\*\* that could be causative of sudden death.

\*parents

- \*\*due to ischemic heart disease or sudden cardiac death before 55 years of age (men) or 65 years of age (women)
- \*\*\*such as known coronary artery disease, congestive heart failure, or terminal cancer
- 20. Any clinically significant ECG abnormality, in the opinion of the site investigator, at screening and at admission to the confinement/hospital unit.
- 21. Donation of >500 mL of blood within the 30 days prior to admission to the confinement/hospital unit.
- 22. Plans to donate blood during the study or up to 14 days after dosing.
- 23. Persons with a transjugular intrahepatic portosystemic shunt.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

All participants will receive a single 200 mg tablet of Pretomanid.

## 4.4.2. Identity of Investigational Product(s)

Pretomanid, a nitroimidazooxazine, is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease, which may improve the current high rate of noncompliance for TB treatment. Pretomanid acts by inhibiting *Mycobacterium tuberculosis* cell wall biosynthesis, as well as by generating reactive nitrogen species.

Pretomanid will be provided by the Global Alliance for TB Drug Development according to the terms of the Clinical Trials Agreement between the TB Alliance and NIAID.

For this study, Pretomanid 200 mg tablets are white to off-white, odorless and oval in appearance. Study drug will be packaged in high-density polyethylene (HDPE) bottles, each containing 50 tablets, and in blister-strips comprised of a thermoformable-film and a lidding foil configuration, each strip containing 7 individual tablets. Sites will receive study product in either packaging depending on supply. Study product in either form of packaging should be stored at 15-30°C (59-86°F).

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

There is no randomization performed for this study. Subjects are assigned to the 3 hepatically impaired groups based on the Child-Pugh score, with approximately 6 subjects in each of the hepatic impairment groups (Groups 1, 2, and 3) and approximately 18 non-hepatically impaired subjects in Group 4.

#### 4.4.4. Selection of Doses in the Study

The PK profile for Pretomanid following oral dosing was consistent for healthy subjects and subjects with pulmonary TB. Pretomanid was readily absorbed after oral administration and slowly eliminated in plasma. Pretomanid plasma concentrations increased in a dose-related manner after single-dose administration of up to 1000 mg in healthy subjects and subjects with TB, but the increase was less than dose proportional,

particularly at doses above 200 mg/day. There is a trend towards increased side effects with increasing dosages (8). Furthermore, efficacy studies have shown equivalent early bacterial activity at dosages ranging from 200mg to 1200mg. The doses of Pretomanid that will be evaluated in regimens in Phase 3 are 100 mg and 200 mg. Hence, the dosage of Pretomanid for this study will be 200mg daily.

## 4.4.5. Selection and Timing of Dose for Each Subject

A single 200 mg tablet will be administered orally on the morning of Day 1 with 240 mL of water following an overnight fast. All participants will receive the same study product.

#### 4.4.6. Blinding

Not applicable; this is an open-label study.

## 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines will be recorded on the appropriate data collection form. Concomitant medications recorded will include all current medications and medications taken within 30 days prior to signing the informed consent and during the study period. Medications reported in the electronic case report form (eCRF) are limited to those taken within 30 days prior to the study drug administration through Day 12 of the study. Prescription and over-the-counter drugs will be included as well as herbals, vitamins, and supplements.

Systemic medications that might interfere with the evaluation of the investigational product should not be used unless absolutely necessary. A subject will be withdrawn for use of excluded medications. Medications in this category include the prohibited medications per the Subject Exclusion Criteria (Section 4.3.2). The excluded CYP450 inducers are: Carbemazepines, Rifampicin, Alcohol (of greater than one drink per day or seven drinks per week), Phenytoin, Griseofulvin, Phenobarbital and Sulphonylureas. The excluded CYP450 inhibitors are: Sodium valproate, Isoniazid, Ketoconazole, Fluconazole, Chloramphenicol, Erythromycin, Sulfonamides, Ciprofloxacin, Metronidazole, and grapefruit juice.

#### 4.4.8. Treatment Compliance

All subjects are to receive a single dose of study product administered in the clinic.

# 4.5. Pharmacokinetics and Safety Variables

See Table 3 for a schedule of study procedures.

#### 4.5.1. Pharmacokinetics Variables

- 1. The pharmacokinetics of a single-dose of Pretomanid will be assessed from serial blood samples collected prior to dosing (Day 1 and at multiple time points post dosing: 1 h, 2 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h, and 96 h. The primary outcome measure will be total plasma concentration of Pretomanid. The following will be determined:
  - a.  $AUC_{(0-\infty)}$ : Area under the concentration time-curve extrapolated to infinity
  - b.  $AUC_{(0-last)}$ : Area under the concentration time-curve to the last concentration above the lower limit of quantitation
  - c. C<sub>max</sub>: Maximum Pretomanid concentration
  - d. T<sub>max</sub>: Time of maximum Pretomanid concentration

- e.  $t_{(1/2)}$ : Apparent terminal elimination half-life
- f. CL/F: Apparent oral clearance calculated from Dose/AUC<sub>(0-∞)</sub>
- g. V<sub>d</sub>/F: Apparent Volume of Distribution

## 4.5.2. Safety Variables

- 1. The secondary outcome measures will be:
  - a. Incidence and severity serious adverse events reported at any time from the time of study treatment through the end of the study.
  - b. Incidence and severity of related adverse events reported at any time from the time of study treatment through Day 12.
  - c. Summary of physical examination findings (height at baseline, and weight at serial time points from Day of Admission until Day 12), vital signs (serial time points from Day of Admission until Day 12), safety laboratory parameters (Day of Admission, as well as Days 2, 5, and 12), and ECG data (Day of Admission and Day 12).

## 5. SAMPLE SIZE CONSIDERATIONS

The sample size was determined based on feasibility and FDA guidance (12). Following FDA guidance, enrollment is anticipated to include at least 6 subjects in each arm. This sample size is expected to estimate the group differences with adequate precision. Previous studies of Pretomanid have estimated coefficients of variation (CV) of <21% after 250 mg dosing (N=8) and <33% after 200 mg dosing (N=6) for single dose  $AUC_{(0-\infty)}$  and  $C_{max}$  in healthy adult subjects (11). Assuming an observed two-fold difference between the group with severe hepatic impairment and matched controls with no correlation between matched pairs and a coefficient of variation of 25%, a 90% confidence interval for the fold difference between severely impaired and non-hepatically impaired group is (1.55, 2.59).

#### 6. GENERAL STATISTICAL CONSIDERATIONS

## **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by impairment group and subject, and when appropriate by visit number within subject. In general, the last recorded value prior to study drug administration will be considered as baseline. All summary tables will be structured with a column for each impairment group in the order (Mild Hepatic Impairment, Moderate Hepatic Impairment, Severe Hepatic Impairment, Matched Controls) and will be annotated with the total population size relevant to that table/impairment group, including any missing observations. More details will be provided for reporting pharmacokinetic results in Section 10.

## **6.2.** Timing of Analyses

Two SMC interim safety reviews are planned.

- 1. After 3 subjects with mild hepatic impairment are enrolled and completed follow-up through Day 12. This review will be completed prior to opening enrollment for subjects with moderate or severe hepatic impairment. Enrollment of subjects with mild hepatic impairment and matched controls may continue during the safety review.
- 2. After 3 subjects with moderate or severe hepatic impairment are enrolled and complete follow-up through Day 12. Enrollment of subjects with mild hepatic impairment, moderate hepatic impairment, severe hepatic impairment, and matched controls may continue during the safety review.

Each interim safety review will present data by impairment group including AEs, SAEs, clinical laboratory tests, vital signs, PK analysis and 12-lead ECG. Cumulative data for all subjects enrolled will be included in the safety reviews.

Interim safety reviews will not include any statistical hypothesis testing.

The final analysis will be performed after database lock.

# **6.3.** Analysis Populations

Summaries and analysis of safety data will be presented for the Safety Population. Summaries and analysis of pharmacokinetics data will be presented for the Pharmacokinetics Population. A tabular listing of all subjects, visits, and observations excluded from the analysis populations will be provided in the CSR (Table 7; Listing 1; and Listing 4).

#### **6.3.1.** Safety Population

The safety analysis set will include all participants who receive study product.

## 6.3.2. Pharmacokinetics Population

The PK analysis set will consist of participants in the safety population who have evaluable plasma PK samples for the estimation of  $C_{max}$  or AUC  $(0-\infty)$ . Subjects may also be excluded from analysis for reasons such

as wrong dose or eating before a dose. What constitutes a reason for exclusion will be assessed on a case-by-case basis by DMID and the VTEU PI.

## 6.4. Covariates and Subgroups

This study is not powered for formal subgroup analyses and none will be explored.

## 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier.

## 6.6. Interim Analyses and Data Monitoring

See Section 6.2.

#### 6.7. Multicenter Studies

This study will take place at two VTEU sites, Duke University and St. Louis University. Data will be pooled across both clinical sites except for demographics which will be summarized by site and the comparison of PK parameters will be presented according to site and impairment group (if applicable, as described in Section 10.3).

## 6.8. Multiple Comparisons/Multiplicity

This study was designed to test the hypothesis that Pretomanid PK parameters following drug exposure will differ between patients with hepatic impairment and non-hepatically impaired controls. This results in three comparisons, however no adjustment for multiple comparisons is planned.

## 7. STUDY SUBJECTS

## 7.1. Disposition of Subjects

Table 8 will present a summary of the reasons that subjects were screened but not enrolled.

The composition of analysis populations, including reasons for subject exclusion, by impairment group, is presented in Table 7.

The disposition of subjects in the study will be tabulated by impairment group (Table 6). The table shows the total number of subjects screened, enrolled, who received treatment, completed all hourly assessments, and the number who completed the Day 12 follow-up.

A flowchart showing the disposition of study subjects, adapted from the Consort Statement (12) will be included (Figure 1). This figure will present the number of subjects screened, enrolled, terminated early, and analyzed, by impairment group.

A listing of subjects who are terminated from study follow-up and the reason will be included in Listing 1.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and impairment group for all subjects (Table 4). All subject-specific protocol deviations and non-subject specific protocol deviations will be included in Appendix 3 as data listings (Listing 2 and Listing 3, respectively).

# 8. EFFICACY EVALUATION

This study is primarily a pharmacokinetics study and does not include an efficacy evaluation.

## 9. SAFETY EVALUATION

All summaries and analysis of safety data will be presented for the Safety Analysis Population. Safety summaries will be presented overall and by impairment group.

Listings will be sorted by impairment group, subject ID, parameter (if applicable), and visit (if applicable).

Continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. All categorical measures will be summarized by the frequency and percentages (based on the non-missing sample size) of observed levels. The denominator for the percentages may be based on the number of non-missing observations for an assessment or based on the number of subjects in a population. This will be described for each table.

## 9.1. Demographic and Other Baseline Characteristics

Summaries of age, height, weight (measured at screening), sex, ethnicity, and race will be presented by impairment group and overall (Table 11; Table 12) as well as by site (Table 9 and Table 10). Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option.

Individual subject listings (Appendix 3) will be presented for all demographics (Listing 5).

#### 9.1.1. Prior and Concurrent Medical Conditions

Complete medical history will be obtained by interview of subjects at the screening visit and will be reviewed and/or updated on Day 1 prior to dosage. Subjects will be queried regarding a history of significant medical disorders of the head, eyes, ears, nose, throat, mouth, cardiovascular system, lungs, gastrointestinal tract, liver, pancreas, kidney, urologic system, nervous system, blood, lymph nodes, endocrine system, musculoskeletal system, skin, and genital/reproductive tract. A history of any allergies, cancer, immunodeficiency, psychiatric illness, substance abuse, and autoimmune disease will be solicited.

All current illnesses and pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 21.0 or higher. Summaries of subjects' pre-existing medical conditions will be presented by impairment group (Table 13).

Individual subject listings will be presented for all medical conditions (Listing 6).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by WHO Drug Terms 2 and 3 and impairment group (Table 140).

Individual subject listings will be presented for all concomitant medications (Listing 14).

# **9.2.** Measurements of Treatment Compliance

Any subjects who were enrolled but not dosed will be presented by impairment group as part of the subject disposition table (Table 6).

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the total population size. All adverse events reported will be included in the summaries and analyses. Adverse event grading scales are presented in Table 5.

An overall summary of adverse events is presented in Table 14.

#### 9.3.1. Unsolicited Adverse Events

The proportion of subjects reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term for each impairment group. Denominators for percentages are the number of subjects who received Pretomanid being summarized.

Adverse events by subject will be presented in Listing 7.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, and impairment group:

- Subject incidence and total frequency of adverse events over time by dose with 95% CI (Days 1-5, Days > 5) (Table 15; Table 16; Table 17; and Table 18);
- Summary of severity and relationship to study product (Table 19);
- Subject listing of non-serious adverse events of moderate or greater severity (Table 21);
- Bar chart of serious and non-serious related adverse events by severity and MedDRA system organ class (Figure 3 and Figure 4).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Adverse Event Description, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

• Deaths and Serious Adverse Events (Table 20).

# 9.5. Pregnancies

Pregnancy is not considered an adverse event; however, for females, information will be collected for any pregnancies which occur during study drug administration until the Study Day 12 Visit. Male subjects should notify the study team if a pregnancy occurs in a partner within 3 months after study drug administration. If the male subject reports a pregnancy, information about complications during pregnancy, labor and delivery, or congenital birth defects will be collected from the male subject's female partner using a site-specific Pregnant Partner Information and Authorization form. Certain pregnancy outcomes (congenital anomaly or birth defect in an offspring of a subject taking study drug) will require submission as an SAE. A listing of pregnancies will be presented (Listing 15; Listing 16; Listing 17; Listing 18; and Listing 19).

## 9.6. Clinical Laboratory Evaluations

Clinical safety laboratory adverse events will be collected at the time of dosage, at 36 hours post dose (Day 2), Day 5 and Day 12. Chemistry parameters to be evaluated include: total bilirubin, serum albumin, potassium, magnesium, calcium, serum creatinine, blood urea nitrogen (BUN), alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST). For patients with severe hepatic impairment an ammonia level will be drawn at screening and will be used as a baseline reading for safety purposes, not as a study entry criterion. Hematology parameters to be evaluated included: hematocrit, hemoglobin, red blood cell count, white blood cell count, automated differential (absolute neutrophils, absolute eosinophils, absolute basophils, absolute lymphocytes, absolute monocytes), and platelet count. The coagulation parameter international normalized ratio (INR) is to be evaluated. Urinalysis parameters to be evaluated by dipstick include: protein, glucose and blood. If any of the urinalysis parameters are positive by dipstick then the sample will be analyzed by reflex microscopy and the results for protein, glucose and blood will be summarized. Grading scales for safety laboratory parameters are presented in Table 5.

The number and percentage of subjects with at least one clinical safety laboratory of mild or greater severity through Day 12 is presented in the overall summary of adverse events (Table 14).

The distribution of chemistry results by severity, time point, and impairment group will be presented beginning at Table 26 and concluding at Table 47. The distribution of hematology results by severity, time point, and impairment group will be presented beginning at Table 58 and concluding at Table 79. The distribution of urine dipstick results by timepoint and impairment group will be shown in Table 90. The distribution of urinalysis results by severity, time point, and impairment group will be presented in Table 91; Table 92; Table 93; Table 94; Table 95; Table 96; Table 97; and Table 98. The distribution of coagulation results by severity, time point, and impairment group will be presented in Table 102 and Table 103. Descriptive statistics including mean, standard deviation, median, minimum and maximum values by time point, for each laboratory parameter, will be summarized in Table 48 and concluding at Table 57 (chemistry); Table 80 and concluding at Table 89 (hematology); Table 99 (Urinalysis); and Table 104 (Coagulation). Table 100; and Table 101 will show distribution of categorical urinalysis results. Shift tables will be presented for each laboratory parameter beginning at Table 105 and concluding at Table 128. Change from baseline plots for continuous laboratory parameters will also be presented beginning at Figure 5 and concluding with Figure 25.

Listing 8; Listing 9; Listing 10; and Listing 11 will provide complete listings of individual clinical laboratory results with applicable reference ranges. Table 22; Table 23; Table 24; and Table 25 will provide listings of abnormal laboratory values.

# 9.7. Vital Signs and Physical Evaluations

Vital sign measurements included oral temperature, pulse, systolic blood pressure, and diastolic blood pressure. Vital signs will be summarized at admission (Day -1), Day 1 pre-dose (Baseline), 1-hour post-dose, 2 hours post-dose, 4 hours post-dose, 5 hours post-dose, 6 hours post-dose, 8 hours post-dose, 12 hours post-dose, 16 hours post-dose, 24 hours post-dose, 36 hours post-dose, Day 3, Day 4, Day 5 and Day 12. Vital signs will be tabulated by visit and impairment group (Table 129 through Table 137; and Listing 12).

Physical Examinations performed at admission and Day 12. The following body systems will be assessed: Abdomen, Cardiovascular/heart Extremities, General Appearance, HEENT, Lymph nodes, Musculoskeletal, Neck, Neurological, Pulmonary/Chest, and Skin (Listing 13). A summary of abnormal physical exam findings

will be shown in Table 138. Weight will be summarized at admission (Day -1), Day 1 pre-dose (Baseline), 1-hour post-dose, 2 hours post-dose, 4 hours post-dose, 5 hours post-dose, 6 hours post-dose, 8 hours post-dose, 12 hours post-dose, 16 hours post-dose, 24 hours post-dose, 36 hours post-dose, Day 3, Day 4, Day 5 and Day 12. Weight will be tabulated by visit and impairment group (Table 139).

#### 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 14). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and impairment group for the Safety population (Table 140).

## 9.9. Other Safety Measures

ECG intervals (RR, QRS, QT, QTcF, PR and ventricular rate) will be summarized at the day of admission and Day 12 using descriptive statistics (Table 141; Table 142; Table 143; Table 144; Table 145; and Table 146). The proportion of subjects with bradycardia, tachycardia, conduction system disease (e.g., prolongation of the PR Interval, bundle branch block, fascicular block), arrhythmia (e.g., atrial fibrillation, atrial flutter, premature atrial/ventricular contractions, ventricular tachycardia), and Brugada pattern will be summarized by hepatic impairment group (Table 147). Individual overall interpretation and comments will be provided in Listing 20. Individual ECG interval measurements will be provided in Listing 21.

## 10. PHARMACOKINETICS

Pharmacokinetic (PK) analyses will be performed using noncompartmental analysis (NCA). PK concentrations and noncompartmental parameters will be summarized by impairment group. Statistics include the arithmetic mean, geometric mean (GM), standard deviation (SD), coefficient of variation (CV), minimum (min), maximum (max), and median. PK parameters (AUC<sub>0-last</sub>, AUC<sub>0-\infty</sub>, and C<sub>max</sub>) will be compared between impairment groups using ANOVA models with or without random effects. T<sub>max</sub> will be compared using 90% confidence intervals calculated using the inverted rank score method. Concentrations below the quantitation limit (BQL) prior to first measurable concentration will be imputed as zero.

## 10.1. Summary of Pharmacokinetic Sampling and Sample Properties

Samples with bioanalytical errors reported by the laboratory will be excluded. Collection times of samples missing the actual collection time will be imputed using the nominal collection time. Such samples will be identified in the analysis report (Listing 22).

## 10.2. Pharmacokinetic Analysis

#### **10.2.1.** Concentration Summaries

Drug plasma concentrations will be listed by impairment group, and subject, out of sample time window, and PK analyses-excluded samples indicated (Listing 22). The listings will also indicate the nominal and actual time associated with the sample (nominal time is defined as the time in hours since the first dose).

Potentially important bioanalytical errors and their effect on the PK analysis will be discussed.

Plasma drug concentrations will also be summarized by impairment group (Table 148; Table 149; Table 150; and Table 151) and plotted.

- Figure 26; Figure 27; Figure 28; and Figure 29 (linear) and Figure 33; Figure 34; Figure 35; and Figure 36 (semilogarithmic) will plot all subject plasma PK profiles together by impairment group, as linear and semilogarithmic plots.
- Linear plots of subjects with hepatic impairment with their matched control (Figure 30; Figure 31; and Figure 32).
- Linear plots of plasma mean concentration curves will be shown in Figure 37, with error bars representing +/- 1 standard deviation.
- Semi-logarithmic plots of geometric mean plasma concentration curves will be shown in Figure 38.

#### 10.2.2. Pharmacokinetic Parameters

NCA PK parameters will be calculated using actual post-dose time. Samples with concentrations greater than the LLOQ will be considered for the estimation of  $\lambda_z$ . This slope will be computed from log-transformed concentration data. The correlation between time and concentration in the time points used to estimate  $\lambda_z$  should be sufficiently high ( $R_{adjusted}^2 > 0.9$  for  $\lambda_z$ . to be estimated reliably. At least three samples will be used for the calculation of  $\lambda_z$ . The range of selected time points should include all timepoints post 12 hours inclusive if appropriate.

Samples used to calculate  $\lambda_z$  along with the number of samples used for the calculation will be included in subject listings (Listing 22).

The AUC will be computed using the linear-up log-down (linear-log) trapezoidal method in WinNonlin (Pharsight Corporation, Cary, NC).

All PK parameters will also be summarized by impairment group using descriptive statistics (Table 152; Table 153; Table 154; and Table 155). Additionally, subject-level PK parameters will be presented by participant in the table in the final report.

The following parameters will be estimated:  $C_{max}$ ,  $T_{max}$ ,  $t_{(1/2)}$ ,  $AUC_{(0-last)}$ ,  $AUC_{(0-\infty)}$ , CL/F and  $V_d/F$ . See Section 3.3 for parameter definitions.

## 10.3. Comparison of Impairment Groups

If at least one matching participant in the healthy volunteer group is available in the impairment groups, the following random effects ANOVA model will be used to test for a group by site interaction and if significant (p<0.10), estimate group and site level parameters and compare impairment groups for primary PK parameters:

$$Y_{ij} = \mu + \tau_{[ij]} + \alpha_i + \gamma_k + \tau_{[ij]}\gamma_k + \varepsilon_{ij}.$$

Here, *i* represents the matched block, *j* represents the participant in matched block *i*,  $Y_{ij}$  is the log-transformed PK parameter for participant *j* in block *i*,  $\tau_{[ij]}$  is the impairment group effect for the group in which participant *j* in block *i* belongs,  $\alpha_i$  is the random group effect for matched block *i*,  $\gamma_k$  is the indicator variable for the fixed effect of study site *k*, and  $\tau_{[ij]}\gamma_k$  is the interaction between subject impairment group and site. If no matching participants are available with PK parameters, the standard fixed effects ANOVA model without random effect  $\alpha_i$  will be used. The following SAS code may be used to estimate the model above:

```
proc mixed data=impairment;
class match group (ref="Matched Control") site;
model logPKpar = group site group*site / solution cl alpha=0.10;
random match;
lsmeans group site group*site;
run:.
```

The estimates from this model can be exponentiated to get fold differences.

If the group by site interaction is not significant then the following model will be used to estimate group level parameters:

$$Y_{ij} = \mu + \tau_{[ij]} + \alpha_i + \gamma_k + \varepsilon_{ij}$$

The following SAS code may be used to estimate the model above:

```
proc mixed data=impairment;
class match group (ref="Matched Control") site;
model logPKpar = group site / solution cl alpha=0.10;
random match;
lsmeans group;
```

run;.

The estimates from this model can be exponentiated to get fold differences.

Pairwise fold differences in drug exposure will be calculated to compare each of the mild, moderate, and severe impairment groups with non-hepatically impaired controls. Fold difference and mean will be estimated by ANOVA and shown using 90% confidence intervals. An adjustment to the confidence level for multiple comparisons is not planned (Table 156).

 $T_{max}$  will be summarized in each impairment group using the median, and group differences will be assessed using nonparametric confidence intervals computed using the inverted rank score method (Table 157). Medians and confidence intervals will also be computed for each site. If the confidence intervals do not overlap between sites, then the  $T_{max}$  will also be summarized by site.

Summary box plots of PK parameters by impairment group (and site if appropriate) will also be prepared (Figure 39; Figure 40; Figure 41; Figure 42; Figure 43; and Figure 44).

# 11. IMMUNOGENICITY

Not applicable.

# 12. OTHER ANALYSES

Not Applicable.

## 13. REPORTING CONVENTIONS

P-values  $\geq$ 0.001 and  $\leq$ 0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001" The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but <1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures. Drug concentrations, AUCs, and  $C_{max}$  and their summary statistics will have the same number of significant digits as the drug concentrations reported by the bioanalytical laboratory. Other PK parameters will be reported to 1 decimal place.
#### 14. TECHNICAL DETAILS

Estimation of NCA parameters will be performed in a validated version of WinNonlin version 6.3 or later, or a similar software package. WinNonlin, SAS version 9.3 or later or R statistical computing software 3.4.2 or higher will be used to generate all tables, figures, and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

No changes in the conduct of the study or planned analysis.

#### 16. REFERENCES

- 1. ICH. International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Efficacy Guidelines. Available from:

  <a href="https://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">https://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>;

  The state of the st
  - E3: https://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E3/E3\_Guideline.pdf;
  - E8: https://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E8/Step4/E8\_Guideline.pdf;
  - E9: https://www.ich.org/fileadmin/Public Web Site/ICH Products/Guidelines/Efficacy/E9/Step4/E9 Guideline.pdf
- 2. Organization WH. Global Tuberculosis Report2016.
- 3. Murray CJ, Ortblad KF, Guinovart C, Lim SS, Wolock TM, Roberts DA, Dansereau EA, Graetz N, Barber RM, Brown JC, Wang H, Duber HC, Naghavi M, Dicker D, Dandona L, Salomon JA, Heuton KR, Foreman K, Phillips DE, Fleming TD, Flaxman AD, Phillips BK, Johnson EK, Coggeshall MS, Abd-Allah F, Abera SF, Abraham JP, Abubakar I, Abu-Raddad LJ, Abu-Rmeileh NM, Achoki T, Adeyemo AO, Adou AK, Adsuar JC, Agardh EE, Akena D, Al Kahbouri MJ, Alasfoor D, Albittar MI, Alcala-Cerra G, Alegretti MA, Alemu ZA, Alfonso-Cristancho R, Alhabib S, Ali R, Alla F, Allen PJ, Alsharif U, Alvarez E, Alvis-Guzman N, Amankwaa AA, Amare AT, Amini H, Ammar W, Anderson BO, Antonio CA, Anwari P, Arnlov J, Arsenijevic VS, Artaman A, Asghar RJ, Assadi R, Atkins LS, Badawi A, Balakrishnan K, Banerjee A, Basu S, Beardsley J, Bekele T, Bell ML, Bernabe E, Beyene TJ, Bhala N, Bhalla A, Bhutta ZA, Abdulhak AB, Binagwaho A, Blore JD, Basara BB, Bose D, Brainin M, Breitborde N, Castaneda-Orjuela CA, Catala-Lopez F, Chadha VK, Chang JC, Chiang PP, Chuang TW, Colomar M, Cooper LT, Cooper C, Courville KJ, Cowie BC, Criqui MH, Dandona R, Dayama A, De Leo D, Degenhardt L, Del Pozo-Cruz B, Deribe K, Des Jarlais DC, Dessalegn M, Dharmaratne SD, Dilmen U, Ding EL, Driscoll TR, Durrani AM, Ellenbogen RG, Ermakov SP, Esteghamati A, Faraon EJ, Farzadfar F, Fereshtehnejad SM, Fijabi DO, Forouzanfar MH, Fra Paleo U, Gaffikin L, Gamkrelidze A, Gankpe FG, Geleijnse JM, Gessner BD, Gibney KB, Ginawi IA, Glaser EL, Gona P, Goto A, Gouda HN, Gugnani HC, Gupta R, Hafezi-Nejad N, Hamadeh RR, Hammami M, Hankey GJ, Harb HL, Haro JM, Havmoeller R, Hay SI, Hedayati MT, Pi IB, Hoek HW, Hornberger JC, Hosgood HD, Hotez PJ, Hoy DG, Huang JJ, Iburg KM, Idrisov BT, Innos K, Jacobsen KH, Jeemon P, Jensen PN, Jha V, Jiang G, Jonas JB, Juel K, Kan H, Kankindi I, Karam NE, Karch A, Karema CK, Kaul A, Kawakami N, Kazi DS, Kemp AH, Kengne AP, Keren A, Kereselidze M, Khader YS, Khalifa SE, Khan EA, Khang YH, Khonelidze I, Kinfu Y, Kinge JM, Knibbs L, Kokubo Y, Kosen S, Defo BK, Kulkarni VS, Kulkarni C, Kumar K, Kumar RB, Kumar GA, Kwan GF, Lai T, Balaji AL, Lam H, Lan Q, Lansingh VC, Larson HJ, Larsson A, Lee JT, Leigh J, Leinsalu M, Leung R, Li Y, De Lima GM, Lin HH, Lipshultz SE, Liu S, Liu Y, Lloyd BK, Lotufo PA, Machado VM, Maclachlan JH, Magis-Rodriguez C, Majdan M, Mapoma CC, Marcenes W, Marzan MB, Masci JR, Mashal MT, Mason-Jones AJ, Mayosi BM, Mazorodze TT, McKay AC, Meaney PA, Mehndiratta MM, Mejia-Rodriguez F, Melaku YA, Memish ZA, Mendoza W, Miller TR, Mills EJ, Mohammad KA, Mokdad AH, Mola GL, Monasta L, Montico M, Moore AR, Mori R, Moturi WN, Mukaigawara M, Murthy KS, Naheed A, Naidoo KS, Naldi L, Nangia V, Narayan KM, Nash D, Nejjari C, Nelson RG, Neupane SP, Newton CR, Ng M, Nisar MI, Nolte S, Norheim OF, Nowaseb V, Nyakarahuka L, Oh IH, Ohkubo T, Olusanya BO, Omer SB, Opio JN, Orisakwe OE, Pandian JD, Papachristou C, Caicedo AJ, Patten SB, Paul VK, Pavlin BI, Pearce N, Pereira DM, Pervaiz A, Pesudovs K, Petzold M, Pourmalek F, Qato D, Quezada AD, Quistberg DA, Rafay A, Rahimi K, Rahimi-Movaghar V, Ur Rahman S, Raju M, Rana SM, Razavi H, Reilly RQ, Remuzzi G, Richardus JH, Ronfani L, Roy N, Sabin N, Saeedi MY, Sahraian MA, Samonte GM, Sawhney M, Schneider IJ, Schwebel DC, Seedat S,

Sepanlou SG, Servan-Mori EE, Sheikhbahaei S, Shibuya K, Shin HH, Shiue I, Shivakoti R, Sigfusdottir ID, Silberberg DH, Silva AP, Simard EP, Singh JA, Skirbekk V, Sliwa K, Soneji S, Soshnikov SS, Sreeramareddy CT, Stathopoulou VK, Stroumpoulis K, Swaminathan S, Sykes BL, Tabb KM, Talongwa RT, Tenkorang EY, Terkawi AS, Thomson AJ, Thorne-Lyman AL, Towbin JA, Traebert J, Tran BX, Dimbuene ZT, Tsilimbaris M, Uchendu US, Ukwaja KN, Uzun SB, Vallely AJ, Vasankari TJ, Venketasubramanian N, Violante FS, Vlassov VV, Vollset SE, Waller S, Wallin MT, Wang L, Wang X, Wang Y, Weichenthal S, Weiderpass E, Weintraub RG, Westerman R, White RA, Wilkinson JD, Williams TN, Woldeyohannes SM, Wong JQ, Xu G, Yang YC, Yano Y, Yentur GK, Yip P, Yonemoto N, Yoon SJ, Younis M, Yu C, Jin KY, El Sayed Zaki M, Zhao Y, Zheng Y, Zhou M, Zhu J, Zou XN, Lopez AD, Vos T. Global, regional, and national incidence and mortality for HIV, tuberculosis, and malaria during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014;384(9947):1005-70. Epub 2014/07/26. doi: 10.1016/S0140-6736(14)60844-8

S0140-6736(14)60844-8 [pii]. PubMed PMID: 25059949.

- 4. Organization WH. Global tuberculosis report (2012). Geneva, Switzerland: 2012.
- 5. Comstock GW. Epidemiology of tuberculosis. Am Rev Respir Dis. 1982;125(3 Pt 2):8-15. Epub 1982/03/01. PubMed PMID: 7073104.
- 6. Maggi N, Pasqualucci CR, Ballotta R, Sensi P. Rifampicin: a new orally active rifamycin. Chemotherapy. 1966;11(5):285-92. Epub 1966/01/01. PubMed PMID: 5958716.
- 7. Organization WH. Treatment of tuberculosis. Guidelines for national programmes, 3rd ed. Geneva, Switzerland 2003. Available from: http://www.who.int/tb/publications/2008/en/index.html.
- 8. Diacon AH, Dawson R, Hanekom M, Narunsky K, Maritz SJ, Venter A, Donald PR, van Niekerk C, Whitney K, Rouse DJ, Laurenzi MW, Ginsberg AM, Spigelman MK. Early bactericidal activity and pharmacokinetics of PA-824 in smear-positive tuberculosis patients. Antimicrob Agents Chemother. 2010;54(8):3402-7. Epub 2010/05/26. doi: 10.1128/AAC.01354-09
  - AAC.01354-09 [pii]. PubMed PMID: 20498324; PMCID: 2916303.
- 9. Chang KC, Leung CC, Yew WW, Chan SL, Tam CM. Dosing schedules of 6-month regimens and relapse for pulmonary tuberculosis. Am J Respir Crit Care Med. 2006;174(10):1153-8. Epub 2006/08/16. doi: 200605-637OC [pii]
  - 10.1164/rccm.200605-637OC. PubMed PMID: 16908866.
- 10. Kruk ME, Schwalbe NR, Aguiar CA. Timing of default from tuberculosis treatment: a systematic review. Trop Med Int Health. 2008;13(5):703-12. Epub 2008/02/13. doi: 10.1111/j.1365-3156.2008.02042.x
  - TMI2042 [pii]. PubMed PMID: 18266783.
- 11. Caminero JA, Sotgiu G, Zumla A, Migliori GB. Best drug treatment for multidrug-resistant and extensively drug-resistant tuberculosis. Lancet Infect Dis. 2010;10(9):621-9. Epub 2010/08/28. doi: 10.1016/S1473-3099(10)70139-0
  - S1473-3099(10)70139-0 [pii]. PubMed PMID: 20797644.

- 12. FDA. Guidance for Industry: Pharmacokinetics in Patients with Impaired Hepatic Function: Study Design, Data Analysis, and Impact on Dosing and Labeling. 2003. Available from: <a href="http://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm072123.pdf">http://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm072123.pdf</a>
- 13. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.

#### 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

## **APPENDICES**

## APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Study Design |
|---|---|
| Table 2: | Summary of 4 Pretomanid Phase 2 studies |
| Table 3: | Schedule of Study Procedures |
| Table 4: | Distribution of Protocol Deviations by Category, Type, and Impairment Group47 |
| Table 5: | Laboratory/Clinical Adverse Event Grading Scale |
| Table 6: | Subject Disposition by Impairment Group |
| Table 7: | Analysis Populations by Impairment Group53 |
| Table 8: | Ineligibility Summary of Screen Failures |
| Table 9: | Summary of Categorical Demographic and Baseline Characteristics by Site56 |
| Table 10: | Summary of Continuous Demographic and Baseline Characteristics by Site57 |
| Table 11: | Summary of Categorical Demographic and Baseline Characteristics by Impairment Group |
| Table 12: | Summary of Continuous Demographic and Baseline Characteristics by Impairment Group |
| Table 13: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Impairment Group |
| Table 14: | Overall Summary of Adverse Events |
| Table 15: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group – Mild Hepatic Impairment |
| Table 16: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group – Moderate Hepatic Impairment |
| Table 17: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group – Severe Hepatic Impairment |
| Table 18: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group – Matched Controls |
| Table 19: | Incidence of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Impairment Group |
| Table 20: | Listing of Serious Adverse Events |
| Table 21: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events67 |
| Table 22: | Listing of Abnormal Laboratory Results - Chemistry |
| Table 23: | Listing of Abnormal Laboratory Results - Hematology69 |
| Table 24: | Listing of Abnormal Laboratory Results - Urinalysis |
| Table 25: | Listing of Abnormal Laboratory Results - Coagulation |

| Table 26: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Chemistry Parameter |
|---|---|
| Table 27: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group — Total Bilirubin |
| Table 28: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group — Serum Albumin |
| Table 29: | Chemistry Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – Potassium |
| Table 30: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Magnesium |
| Table 31: | Chemistry Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – Calcium |
| Table 32: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group — Serum Creatinine |
| Table 33: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group - BUN |
| Table 34: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Alkaline Phosphatase |
| Table 35: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group - ALT |
| Table 36: | Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – AST |
| Table 37: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Any Chemistry Parameter82 |
| Table 38: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Total Bilirubin83 |
| Table 39: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Serum Albumin83 |
| Table 40: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Range,<br>Maximum Severity, Time Point, and Impairment Group – Potassium84 |
| Table 41: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Magnesium |
| Table 42: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Range, Maximum Severity, Time Point, and Impairment Group – Calcium87 |
| Table 43: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Serum Creatinine88 |

| Table 44: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – BUN |
|---|---|
| Table 45: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Alkaline Phosphatase90 |
| Table 46: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – ALT90 |
| Table 47: | Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – AST90 |
| Table 48: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Total Bilirubin (mg/dL) |
| Table 49: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Serum Albumin (g/dL) |
| Table 50: | Chemistry Laboratory Summary Statistics by Range, Time Point, and Impairment Group – Potassium (mmol/dL) |
| Table 51: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Magnesium (mg/dL) |
| Table 52: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Calcium (mg/dL) |
| Table 53: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Serum Creatinine (mg/dL) |
| Table 54: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – BUN (mg/dL) |
| Table 55: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Alkaline Phosphatase (U/L) |
| Table 56: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – ALT (U/L)92 |
| Table 57: | Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – AST (U/L) |
| Table 58: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment<br>Group – Any Hematology Parameter |
| Table 59: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment<br>Group – Hematocrit |
| Table 60: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment<br>Group – Hemoglobin94 |
| Table 61: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment<br>Group – Red Blood Cell Count94 |

| Table 62: | Hematology Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – White Blood Cell Count95 |
|---|---|
| Table 63: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Neutrophils |
| Table 64: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Eosinophils98 |
| Table 65: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Basophils98 |
| Table 66: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Lymphocytes |
| Table 67: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Monocytes |
| Table 68: | Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Platelets |
| Table 69: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Any Hematology Parameter99 |
| Table 70: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Hematocrit100 |
| Table 71: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Hemoglobin |
| Table 72: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Red Blood Cell Count100 |
| Table 73: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – White Blood Cell Count101 |
| Table 74: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Absolute Neutrophils |
| Table 75: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Absolute Eosinophils104 |
| Table 76: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Absolute Basophils104 |
| Table 77: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Absolute Lymphocytes104 |
| Table 78: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Absolute Monocytes |
| Table 79: | Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Platelets |

| Table 80: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Hematocrit (%) |
|---|---|
| Table 81: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Hemoglobin (g/dL) |
| Table 82: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group $-$ Red Blood Cell Count $(x10^{12}/L)$ |
| Table 83: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – White Blood Cell Count (x10 <sup>9</sup> /L) |
| Table 84: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Neutrophils (x10 <sup>9</sup> /L) |
| Table 85: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Eosinophils (x10 <sup>9</sup> /L) |
| Table 86: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Basophils (x10 <sup>9</sup> /L) |
| Table 87: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Lymphocytes (x10 <sup>9</sup> /L) |
| Table 88: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Monocytes (x10 <sup>9</sup> /L) |
| Table 89: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Platelets (x10 <sup>9</sup> /L) |
| Table 90: | Urinalysis Laboratory Results by Parameter, Time Point, and Impairment Group107 |
| Table 91: | Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Urinalysis Parameter |
| Table 92: | Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group - Protein |
| Table 93: | Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group - Glucose |
| Table 94: | Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group - Urine Blood |
| Table 95: | Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Any Urinalysis Parameter110 |
| Table 96: | Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Protein |
| Table 97: | Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Glucose |

| Table 98: | Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Urine Blood |
|---|---|
| Table 99: | Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Blood (rbc/hpf) |
| Table 100: | Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Protein |
| Table 101: | Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Glucose |
| Table 102: | Coagulation Laboratory Results by Maximum Severity, Time Point, and Impairment Group – INR |
| Table 103: | Abnormal Coagulation Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – INR |
| Table 104: | Coagulation Laboratory Summary Statistics by Time Point and Impairment Group – INR |
| Table 105: | Chemistry Shift Tables by Time Point and Impairment Group – Total Bilirubin121 |
| Table 106: | Chemistry Shift Tables by Time Point and Impairment Group – Serum Albumin121 |
| Table 107: | Chemistry Shift Tables by Time Point and Impairment Group – Potassium121 |
| Table 108: | Chemistry Shift Tables by Time Point and Impairment Group – Magnesium121 |
| Table 109: | Chemistry Shift Tables by Time Point and Impairment Group – Calcium122 |
| Table 110: | Chemistry Shift Tables by Time Point and Impairment Group – Serum Creatinine122 |
| Table 111: | Chemistry Shift Tables by Time Point and Impairment Group – BUN122 |
| Table 112: | Chemistry Shift Tables by Time Point and Impairment Group – Alkaline Phosphatase |
| Table 113: | Chemistry Shift Tables by Time Point and Impairment Group – ALT122 |
| Table 114: | Chemistry Shift Tables by Time Point and Impairment Group – AST122 |
| Table 115: | Hematology Shift Tables by Time Point and Impairment Group – Hematocrit122 |
| Table 116: | Hematology Shift Tables by Time Point and Impairment Group – Hemoglobin122 |
| Table 117: | Hematology Shift Tables by Time Point and Impairment Group – Red Blood Cell Count |
| Table 118: | Hematology Shift Tables by Time Point and Impairment Group – White Blood Cell Count |
| Table 119: | Hematology Shift Tables by Time Point and Impairment Group – Neutrophils122 |
| Table 120: | Hematology Shift Tables by Time Point and Impairment Group – Eosinophils122 |
| Table 121: | Hematology Shift Tables by Time Point and Impairment Group – Basophils122 |

| Table 122: Hematology Shift Tables by Time Point and Impairment Group – Lymphocyte | s122 |
|---|---|
| Table 123: Hematology Shift Tables by Time Point and Impairment Group – Monocytes | 122 |
| Table 124: Hematology Shift Tables by Time Point and Impairment Group – Platelets | 122 |
| Table 125: Coagulation Shift Tables by Time Point and Impairment Group – INR | 122 |
| Table 126: Urinalysis Shift Tables by Time Point and Impairment Group – Protein | 122 |
| Table 127: Urinalysis Shift Tables by Time Point and Impairment Group – Glucose | 122 |
| Table 128: Urinalysis Shift Tables by Time Point and Impairment Group – Blood | 122 |
| Table 129: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Any | |
| Table 130: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Oral Temperature | 126 |
| Table 131: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Pulse | 127 |
| Table 132: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Systo | |
| Pressure | |
| | olic Blood |
| Pressure | olic Blood132 Cemperature |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T | colic Blood<br>132<br>cemperature<br>136 |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T | rolic Blood132 Temperature136141 ic Blood |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T. Table 135: Vital Signs Summary Statistics by Time Point and Impairment Group – Pulse. Table 136: Vital Signs Summary Statistics by Time Point and Impairment Group – Systol | olic Blood132 Semperature136141 ic Blood141 lic Blood |
| Pressure | olic Blood132 Temperature136141 ic Blood141 lic Blood141 |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T. Table 135: Vital Signs Summary Statistics by Time Point and Impairment Group – Pulse Table 136: Vital Signs Summary Statistics by Time Point and Impairment Group – Systol Pressure Table 137: Vital Signs Summary Statistics by Time Point and Impairment Group – Diasto Pressure | colic Blood132 cemperature136141 ic Blood141 lic Blood141142 |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T. Table 135: Vital Signs Summary Statistics by Time Point and Impairment Group – Pulse. Table 136: Vital Signs Summary Statistics by Time Point and Impairment Group – Systol Pressure Table 137: Vital Signs Summary Statistics by Time Point and Impairment Group – Diasto Pressure Table 138: Summary of Abnormal Physical Exam Findings by Impairment Group | colic Blood132 Cemperature136141 ic Blood141 lic Blood141142 eight144 WHO |
| Pressure | colic Blood132 Cemperature136141 ic Blood141 lic Blood141 eight144 WHO150 |
| Pressure | olic Blood132 Semperature136141 ic Blood141 lic Blood141 eight144 WHO150151 |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T Table 135: Vital Signs Summary Statistics by Time Point and Impairment Group – Pulse. Table 136: Vital Signs Summary Statistics by Time Point and Impairment Group – Systol Pressure Table 137: Vital Signs Summary Statistics by Time Point and Impairment Group – Diasto Pressure Table 138: Summary of Abnormal Physical Exam Findings by Impairment Group Table 139: Physical Exam Summary Statistics by Time Point and Impairment Group – Word Table 140: Number and Percentage of Subjects with Prior and Concurrent Medications by Drug Classification and Impairment Group | olic Blood132 Semperature136141 ic Blood141 lic Blood141142 eight144 WHO150151 |
| Pressure Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diast Pressure Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral T. Table 135: Vital Signs Summary Statistics by Time Point and Impairment Group – Pulse. Table 136: Vital Signs Summary Statistics by Time Point and Impairment Group – Systol Pressure Table 137: Vital Signs Summary Statistics by Time Point and Impairment Group – Diasto Pressure Table 138: Summary of Abnormal Physical Exam Findings by Impairment Group – Wordship Time Point and Impairment Group – Wordship Time Point and Impairment Group – Wordship Time Point and Impairment Group – Wordship Time Point and Impairment Group – RR | olic Blood132 demperature136141 dic Blood141 lic Blood141142 deight144 WHO150151151 |
| Pressure | olic Blood132 demperature136141 dic Blood141 lic Blood141142 eight144 deight144 |

| Table 147: | Number and Percentage of Subjects Experiencing ECG Events by Symptom, and Impairment Group |
|---|---|
| Table 148: | Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours) - Mild Hepatic Impairment |
| Table 149: | Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours) - Moderate Hepatic Impairment |
| Table 150: | Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours) - Severe Hepatic Impairment |
| Table 151: | Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours) - Matched Controls |
| Table 152: | Individual and Summary Statistics for Noncompartmental PK Parameters – Mild Hepatic Impairment |
| Table 153: | Individual and Summary Statistics for Noncompartmental PK Parameters – Moderate Hepatic Impairment |
| Table 154: | Individual and Summary Statistics for Noncompartmental PK Parameters – Severe Hepatic Impairment |
| Table 155: | Individual and Summary Statistics for Noncompartmental PK Parameters – Matched Controls |
| Table 156: | Estimated Impairment Group Fold Change for Noncompartmental PK Parameters155 |
| Table 157: | Estimated Impairment Group Shift for Noncompartmental PK Parameters157 |

#### 9.1 Overall Study Design and Plan Description

**Table 1:** Study Design

| Study Group | Severity | N |
|---|---|---|
| Group 1 | Child-Pugh A = 5 to 6 points (Mild Hepatic Impairment) | 6 |
| Group 2 | Child-Pugh B = 7 to 9 points (Moderate Hepatic Impairment) | 6 |
| Group 3 | Child-Pugh C = 10 to 15 points (Severe Hepatic Impairment) | 6 |
| Group 4 | Non-hepatically impaired controls (Matched Controls) | ≤18 |

 Table 2:
 Summary of 4 Pretomanid Phase 2 studies

| Year | N | Pretomanid<br>Regimen | Dosage | Primary<br>Outcome | Mean daily fall in CFU |
|---|---|---|---|---|---|
| 2010 | 60 | Once Daily | 200, 600, 1000,and<br>1200 mg/day | Mean rate of<br>decline in log<br>CFU of TB over<br>14 days | 0.098 (+/-0.072) was equivalent for all four dosages |
| 2012 | 60 | Once Daily | 50, 100, 150, and<br>200 mg/day | Mean rate of<br>decline in log<br>CFU of TB over<br>14 days | $50 mg \ 0.063 \pm 0.058$ $100 mg \ 0.091 \pm 0.073$ $150 mg \ 0.078 \pm 0.074$ $200 mg \ 0.112 \pm 0.070$ |
| 2012 | 81 | Once Daily | Pretomanid + bedaquiline Pretomanid + pyrazinamide Pretomanid + pyrazinamide + moxifloxacin (all Pretomanid dosages were 200mg/day) | Mean rate of<br>decline in log<br>CFU of TB over<br>56 days | Pretomanid+ moxifloxacin+pyrazinamide (0.233) was significantly higher than bedaquiline (0.061), bedaquiline+pyrazinamide (0.131), and comparable with that of standard treatment |
| 2014 | 207 | Once Daily | Pretomanid 200mg + pyrazinamide + moxifloxacin Pretomanid 100mg + pyrazinamide + moxifloxacin Pretomanid 200mg + pyrazinamide + moxifloxacin (Tx MDR-TB) | Mean rate of<br>decline in log<br>CFU of TB over<br>14 days | Pretomanid 200mg + pyrazinamide + moxifloxacin (0.155) Pretomanid 100mg + pyrazinamide + moxifloxacin (0.133) Pretomanid 200mg + pyrazinamide + moxifloxacin (Tx MDR-TB) (0.117) |

#### 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

**Table 3:** Schedule of Study Procedures

| Study Visit | 00A | 00B | 01 | 01A | 01B | 01C | 01D | 01E | 01F | 01G | 01H | 01I | 01J | 02 | 03 | 04 | 05 | Early<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screen<br>-22 to -<br>2 | Admission<br>-1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 3 | 4 | 5 | 12 | |
| Time (Window) | | | (-10 min) | 1 hr<br>(+/-<br>10<br>min) | 2 hr<br>(+/-<br>10<br>min) | 4 hr<br>(+/-<br>10<br>min) | 5 hr<br>(+/-<br>10<br>min) | 6 hr<br>(+/-<br>10<br>min) | 8 hr<br>(+/-<br>10<br>min) | 12 hrs<br>(+/-<br>10<br>min) | 16 hr<br>(+/-<br>10<br>min) | 24 hrs<br>(+/-<br>1 hr) | 36 hrs<br>(+/-<br>1 hr) | 48 hrs<br>(+/-<br>4 hrs) | 72 hrs<br>(+/-<br>4 hrs) | 96 hrs<br>(+/-<br>4 hrs) | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Review Inclusion/<br>Exclusion Criteria | X | X | | | | | | | | | | | | | | | | |
| Demographics <sup>1</sup> | X | | | | | | | | | | | | | | | | | |
| Medical/Surgical<br>History <sup>2</sup> | X | X | | | | | | | | | | | | X | X | X | X | X |
| Physical Examination <sup>3</sup> | X | X | | | | | | | | | | | | | | | X | X |
| Targeted Review of<br>Body Systems <sup>12</sup> | | | | | | | | | | | | | | X | X | X | X | X |
| Concomitant<br>Medication | X | X | | | | | | | | | | | | X | X | X | X | X |
| 12-Lead ECG<br>(Resting) | X | $X^1$ | | | | | | | | | | | | | | | X | |
| Vital Signs <sup>6</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Safety Laboratory Testing (Hematology, Chemistry) <sup>9,11</sup> | $X^4$ | X <sup>13</sup> | | | | | | | | | | | X <sup>10</sup> | | | X | X | |
| Coagulation <sup>9</sup> | $X^4$ | $X^{13}$ | | | | | | | | | | | $X^{10}$ | | | X | X | |
| Urinalysis <sup>9</sup> | X <sup>4</sup> | X <sup>13</sup> | | | | | | | | | | | $X^{10}$ | | | X | X | |
| Pregnancy Test <sup>9</sup> | X <sup>4</sup> | $X^{13}$ | | | | | | | | | | | | | | | X | X |
| Drug and Alcohol<br>Screen <sup>5,8</sup> | X <sup>4</sup> | X | | | | | | | | | | | | | | | | |
| Blood for HIV, HCV,<br>HBsAg testing <sup>8</sup> | X <sup>4</sup> | | | | | | | | | | | | | | | | | |
| Blood for PK<br>Sampling <sup>7</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Discharge from the confinement/hospital unit <sup>14</sup> | | | | | | | | | | | | | X | X | | | | |

**Table 3:** Schedule of Study Procedures (continued)

| Study Visit | 00A | 00B | 01 | 01A | 01B | 01C | 01D | 01E | 01F | 01G | 01H | 01I | 01J | 02 | 03 | 04 | 05 | Early<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screen -22 to - | Admission<br>-1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 3 | 4 | 5 | 12 | |
| Time (Window) | | | (-10 min) | 1 hr<br>(+/-<br>10<br>min) | 2 hr<br>(+/-<br>10<br>min) | 4 hr<br>(+/-<br>10<br>min) | 5 hr<br>(+/-<br>10<br>min) | 6 hr<br>(+/-<br>10<br>min) | 8 hr<br>(+/-<br>10<br>min) | 12 hrs<br>(+/-<br>10<br>min) | 16 hr<br>(+/-<br>10<br>min) | 24 hrs<br>(+/-<br>1 hr) | 36 hrs<br>(+/-<br>1 hr) | 48 hrs<br>(+/-<br>4 hrs) | 72 hrs<br>(+/-<br>4 hrs) | 96 hrs<br>(+/-<br>4 hrs) | | |
| Study Product<br>Administration <sup>7b</sup> | | | X | | | | | | | | | | | | | | | |
| AE Assessment | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| SAE Assessment | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Total blood drawn | 27.5mL | 11.5mL | 6mL | 6mL | 6mL | 6mL | 6mL | 6mL | 6mL | 6mL | 6mL | 6mL | 17.5mL | 6mL | 6mL | 17.5mL | 14.5mL | 0mL |

- 1 Child-Pugh Score calculated for hepatically-impaired subjects at screening
- 2 Complete medical/surgical history taken at screening and interim medical/surgical history as sequent indicated visits.
- 3 Physical examination must include the following organ or body system assessments: skin; head, eyes, ears, nose, and throat; thyroid; neurological; chest and lungs; cardiovascular; abdomen (liver and spleen); lymph nodes; musculoskeletal, and extremities. At early termination visit, a physical examination will be performed.
- 4 If screening laboratory tests are performed within 72 hours of admission to the confinement/hospital unit, the tests do not have to be repeated with the exception of the urine pregnancy test for females of child bearing potential and the urine drug screen for all subjects, which will be repeated.
- 5 Alcohol screen includes alcohol breath test or other suitable test for alcohol (e.g., blood alcohol test).
- 6 Vital sign measurements must include the subject's sitting heart rate, sitting blood pressure (mm Hg), height (screening only), and oral body temperature (°C). Vital signs will be obtained at screening, and on Days -1 to 12 at the following time points:, admission day, prior to dosing, and 30 minutes after dosing, 1, 2, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours and Day 12. Weight will be collected at screening, admission day, prior to dosing, 36, 48, 72, 96 hours and Day 12 time points.

- Blood samples for pharmacokinetic assessments of Pretomanid will be obtained on Days 1 to 5 at the following time points: pre-dose and 1, 2, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose.
- a. The following collection windows are allowed for the PK blood sample time points:
  - i. Pre-dose: -10 minutes
  - ii. Dosing through 16 hours post-dose inclusive:  $\pm 10$  minutes
  - iii. 24 and 36 hours post-dose:  $\pm 1$  hour
  - iv. 48, 72, and 96 hours:  $\pm$  4 hours
- b. Subjects will receive the single oral dose of Pretomanid 200 mg taken with 240 mL of water after overnight fast.
- The following parameters will be used for PK assessments: AUC0-inf, AUC0-t, Cmax, tmax, half-life and CL/F.
- 8 Screening labs include: blood screen for hepatitis B surface antigen (HBsAg) and hepatitis C antibody, alcohol breath test or other suitable test for alcohol (e.g., blood alcohol test), urine screen test for drugs of abuse [amphetamines, barbiturates, benzodiazepines, cocaine metabolites, opiates, cannabinoids, phencyclidine (PCP)] and a blood screen for HIV.

- Safety labs (also performed at screening and 2 hour fasting) include: total bilirubin, serum albumin, electrolytes including potassium, magnesium, and calcium levels, serum creatinine, BUN, alkaline phosphatase, AST, ALT, INR (PT prolongation), CBC w/differential, urinalysis, and pregnancy testing. Pregnancy testing at screening and Day 12 will be serum, and testing at admission will be a urine test.
- 10 Chemistry (2 hour fasting), hematology, coagulation and urinalysis to be done prior to discharge.
- 11 For patients with severe hepatic impairment (Child-Pugh C) an ammonia level will be drawn at screening and will be used as a baseline reading for safety purposes, not as a study entry criterion.
- 12 A targeted review of body systems will be obtained at these visits focused on liver disease and will include questions pertaining to development of ascites, jaundice, pruritis, gastrointestinal bleeding, and encephalopathy. If the subject answers yes to any of these questions, a targeted physical exam will be performed.
- 13 Baseline admissions labs and resting 12-Lead ECG recording may be done within 72 hours of admission or at the time of admission depending on ability to obtain lab results at the site.
- 14 Discharge from confinement/hospital unit either after Visit 01J or Visit 2 depending upon site preference.

#### **10.2** Protocol Deviations

Table 4: Distribution of Protocol Deviations by Category, Type, and Impairment Group

| | | | rment | Moderate<br>Hepatic<br>Impairment<br>(N=X) | | Severe<br>Hepati<br>Impair<br>(N=X) | c | Matched<br>Controls<br>(N=X) | | All Subjects | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No.<br>of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No.<br>of<br>Dev. |
| Eligibility/enrollment | Any type | | | | | | | | | | |
| | Did not meet inclusion criterion | x | x | x | x | | | | | x | x |
| | Met exclusion criterion | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | |
| | Blood not collected | | | | | | | | | | |
| | Urine not collected | | | | | | | | | | |
| | Stool not collected | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | | | |
| | Other | | | | | | | | | | |

Table 4: Distribution of Protocol Deviations by Category, Type, and Treatment Group (continued)

| | | Mild Hepatic<br>Impairment<br>(N=X) | | Moderate<br>Hepatic<br>Impairment<br>(N=X) | | Severe<br>Hepatic<br>Impairment<br>(N=X) | | Matched<br>Controls<br>(N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No.<br>of<br>Subj. | No. of<br>Dev. | | No. of<br>Dev. | No. of<br>Subj. | | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No.<br>of<br>Dev. |
| Treatment administration | Any type | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Note: N= All Enrol | led Subjects | | • | • | • | • | • | | | | • |

# 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

 Table 5:
 Laboratory/Clinical Adverse Event Grading Scale

| Category | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Comments |
|---|---|---|---|---|
| VITAL SIGNS | | | | |
| Fever (°C) ** | 38.0 – 38.4 | 38.5 – 38.9 | ≥ 39.0 | ** Oral temperature; no<br>recent hot or cold<br>beverages or smoking.<br>A protocol should select<br>either °C or °F for<br>inclusion. |
| (°F) ** | 100.4 – 101.1 | 101.2 - 102.0 | ≥ 102.1 | |
| Tachycardia – beats per minute | 101 – 115 | 116 – 130 | > 130 or<br>ventricular<br>dysrhythmias | |
| Bradycardia – beats per minute | 50 – 54 or 45-50<br>bpm if pre-dose<br>visit rate < 60 bpm | 45 – 49 or 40-44<br>if pre-dose visit<br>rate < 60bpm | < 45 or <40bpm if<br>pre-dose visit rate<br><60bpm | |
| Hypertension (systolic) – mm Hg | 141 – 150 | 151 – 160 | > 160 | Assume supine position for 10 min at rest in non-sleeping subjects; for adverse events, need three measurements on the same arm with concordant results. |
| Hypertension (diastolic) – mm Hg | 91 – 95 | 96 – 100 | > 100 | |
| Hypotension (systolic) -mm Hg | 85 – 89 | 80 – 84 | < 80 | |
| Tachypnea – breaths per minute | 23 – 25 | 26 – 30 | > 30 | |
| CARDIOVASCULAR | | | | |
| Arrhythmia | Asymptomatic,<br>transient signs,<br>no Rx required | Recurrent/<br>persistent;<br>symptomatic;<br>Rx required | Unstable<br>dysrhythmia;<br>hospitalization and<br>treatment required | |
| Hemorrhage, Blood Loss | Estimated blood loss ≤ 100 mL | Estimated blood<br>loss > 100 mL,<br>no transfusion<br>required | Transfusion required | |
| QT/QTc prolongation | Male: 441-470 msec | Male: 471-500 msec | > 500 msec<br>OR | |
| | Female:<br>451-470 msec | Female: 471-500 msec: | > 60 msec change<br>from admission visit | |

 Table 5:
 Laboratory/Clinical Event Grading Scale (continued)

| Category | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Comments |
|---|---|---|---|---|
| RESPIRATORY | | | | |
| Cough | Transient- no treatment | Persistent cough; | Interferes with daily activities | |
| Bronchospasm, Acute | Transient; no<br>treatment; 71% -<br>80% FEV1 of peak<br>flow | Requires<br>treatment;<br>normalizes with<br>bronchodilator;<br>FEV1 60% -<br>70% (of peak<br>flow) | No normalization with bronchodilator; FEV1 < 60% of peak flow | |
| Dyspnea | Does not interfere with usual and social activities | Interferes with usual and social activities, no treatment | Prevents daily and usual social activity or requires treatment | |
| GASTROINTESTINAL | | | | |
| Nausea | No interference with activity | Some interference with activity | Prevents daily activities | |
| Vomiting | No interference with activity or 1 – 2 episodes/24 hours | Some interference with activity or > 2 episodes/24 hours | Prevents daily<br>activity or requires<br>IV hydration | |
| Diarrhea | 2 – 3 loose or<br>watery stools or <<br>400 gms/24 hours | 4 – 5 loose or<br>watery stools or<br>400 – 800<br>gms/24 hours | 6 or more loose or<br>watery stools or ><br>800gms/24 hours<br>or requires IV<br>hydration | |
| LABORATORY ADVERSE EV | ENTS | | | |
| Blood, Serum, or Plasma * | | | | |
| Potassium – Hypokalemia mmol/L | 3.1 – <lln< td=""><td>2.7 – 3.0</td><td>&lt;2.7</td><td></td></lln<> | 2.7 – 3.0 | <2.7 | |
| Potassium – Hyperkalemia mmol/L | >ULN - 5.6 | >5.6 - 6.5 | >6.5 | |
| Glucose – Hypoglycemia Fasting – mg/dL # | 61 – <lln< td=""><td>55 – &lt;61</td><td>&lt;55</td><td></td></lln<> | 55 – <61 | <55 | |
| Glucose – Hyperglycemia<br>Fasting – mg/dL # | >ULN – 120 | >120 – 130 | >130 | |
| Blood Urea Nitrogen mg/dL | >ULN – 29 | 30 – 35 | >35 | |
| Creatinine – mg/dL | >ULN – 1.7 | 1.8 - 2.0 | >2.0 | |
| Calcium – hypocalcemia mg/dL | 8.0 – <lln< td=""><td>7.5 – 7.9</td><td>&lt;7.5</td><td></td></lln<> | 7.5 – 7.9 | <7.5 | |

 Table 5:
 Laboratory/Clinical Event Grading Scale (continued)

| Category | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Comments |
|---|---|---|---|---|
| Calcium – hypercalcemia mg/dL | >ULN - 11.0 | 11.1 – 11.5 | >11.5 | |
| Magnesium – hypomagnesemia<br>mg/dL | 1.3 – <lln< td=""><td>1.0 - &lt;1.3</td><td>&lt;1.0</td><td></td></lln<> | 1.0 - <1.3 | <1.0 | |
| Albumin – Hypoalbuminemia g/dL | 2.8 – <lln< td=""><td>2.5 - 2.7</td><td>&lt;2.5</td><td></td></lln<> | 2.5 - 2.7 | <2.5 | |
| Alkaline phosphatase – U/L(Age 18 years) | >ULN - 240 | 241 – 360 | >360 | |
| AST U/L | >ULN - 105 | 106 – 175 | >175 | |
| ALT U/L | >ULN - 105 | 106 – 175 | >175 | |
| Bilirubin (serum total) mg/dL | >ULN - 2.0 | 2.1 – 2.5 | >2.5 | |
| Hemoglobin - g/dL | 10.5 – <lln< td=""><td>9.5 – 10.4</td><td>&lt; 9.5</td><td></td></lln<> | 9.5 – 10.4 | < 9.5 | |
| Hematocrit - % | 32.3 – <lln< td=""><td>28.0 – 32.2</td><td>&lt; 28.0</td><td></td></lln<> | 28.0 – 32.2 | < 28.0 | |
| RBC Decrease (Female) X10^12/L | 3.61 – <lln< td=""><td>3.14 – 3.60</td><td>&lt; 3.14</td><td></td></lln<> | 3.14 – 3.60 | < 3.14 | |
| RBC Decrease (Male)<br>X10E6/uL X10^12/L | 3.89 – <lln< td=""><td>3.28 – 3.88</td><td>&lt; 3.28</td><td></td></lln<> | 3.28 – 3.88 | < 3.28 | |
| WBC Increase X10^9/L | >ULN - 15.0 | 15.1 – 20.0 | > 20.0 | |
| WBC Decrease X10^9/L | 2.5 – <lln< td=""><td>1.5 – 2.4</td><td>&lt; 1.5</td><td></td></lln<> | 1.5 – 2.4 | < 1.5 | |
| Lymphocytes Decrease - X10^9/L | 0.5 – <lln< td=""><td>0.3 - 0.4</td><td>&lt;0.3</td><td></td></lln<> | 0.3 - 0.4 | <0.3 | |
| Neutrophils Decrease - X10^9/L | 1.0 – <lln< td=""><td>0.5 – 1.0</td><td>&lt; 0.5</td><td></td></lln<> | 0.5 – 1.0 | < 0.5 | |
| Monocytes Increased X10^9/L | >ULN - 2.5 | 2.6 – 3.0 | >3.0 | |
| Eosinophils Increased X10^9/L | >ULN - 0.75 | 0.76-1.50 | >1.50 | |
| Basophils Increased X10^9/L | >ULN - 0.40 | 0.41 - 0.80 | >0.80 | |
| Platelets Decreased - X10^9/L | 120 – <lln< td=""><td>100 – 119</td><td>&lt;100</td><td></td></lln<> | 100 – 119 | <100 | |
| INR | >ULN - 1.3 | 1.4 – 1.6 | >1.6 | |
| Urine * | | | | |
| Protein | 1+ | 2+ | > 2+ | |
| Glucose | Trace – 1+ | 2+ | > 2+ | |
| Blood (microscopic) - red blood<br>cells per high power field (rbc/hpf) | 3 – 10 | 11 – 50 | > 50 and/or<br>gross blood | |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters.

<sup>\*</sup> Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

<sup>#</sup>Laboratory Parameter will not be used as halting criteria.

#### 14.1 Description of Study Subjects

#### 14.1.1 Disposition of Subjects

**Table 6:** Subject Disposition by Impairment Group

| Subject | Mild Hepatic<br>Impairment | | Moderate<br>Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment<br>(N=X) | Matched<br>Controls (N=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|
| Disposition | n | % | n | % | | | n | % |
| Screened | | | | | | | X | |
| Enrolled | X | 100 | X | 100 | | | X | 100 |
| Received Treatment | X | xx | X | xx | | | X | xx |
| Completed all hourly assessments | X | xx | x | xx | | | x | xx |
| Completed Follow-up (Study Day 12) <sup>a, b</sup> | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Refer to Listing 16.2.1 for reasons subjects discontinued or terminated early.

Note: N=All Enrolled Subjects

<sup>&</sup>lt;sup>b</sup> Completed all daily assessments following discharge through study day 12.

**Table 7:** Analysis Populations by Impairment Group

| Analysis<br>Populations | | - | | Hepatic<br>Impairment | | | | Matched Controls<br>(N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Excluded | n | % | n | % | n | % | n | % | % | n |
| Safety Population | Any Reason | х | xx | X | xx | | | | | X | XX |
| | Did not receive study product | | | | | | | | | | |
| Pharmacokinetics<br>Population | Any Reason | | | | | | | | | | |
| | Insufficient number of samples for estimation of PK parameters | | | | | | | | | | |
| | Did not meet all inclusion criteria or met exclusion criteria | | | | | | | | | | |

Note: N= Number of subjects enrolled

**Table 8:** Ineligibility Summary of Screen Failures

| Subjects with<br>Hepatic<br>Impairment/<br>Non-Hepatically<br>Impaired Controls | Inclusion/<br>Exclusion<br>Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | <b>%</b> b |
|---|---|---|---|---|
| All Subjects | Inclusion<br>and<br>Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| Subjects with<br>Hepatic Impairment | Inclusion<br>and<br>Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| | Inclusion | Any inclusion criterion | X | xx |
| | | Subject is able to give voluntary written informed consent before any study related procedure is performed | x | xx |
| | | 18-70 years of age, inclusive | X | XX |
| | | (continued) | X | xx |
| | Exclusion | Any exclusion criterion | x | xx |
| | | Hypokalemia (< 3.5mEq/L), severe hypomagnesemia (< 1.1 mg/dL) or severe hypocalcemia (< 7.5 mg/dL) | x | xx |
| | | AST or ALT > 10 times the upper limit of normal | X | XX |
| | | (continued) | x | xx |
| | Eligible but | | | |
| | Not Enrolled | Any Reason | X | XX |
| | | Time Commitment | X | XX |
| | | Concern of Potential Risks | X | XX |
| | | Number of Procedures/Blood Draws | X | XX |
| | | Unable to Contact Subjects | X | XX |
| | | Other | X | XX |
| Non-Hepatically<br>Impaired Controls | Inclusion<br>and<br>Exclusion | Number of subjects failing any eligibility criterion | x | 100 |
| | Inclusion | Any inclusion criterion | x | xx |
| | | Subject is able to give voluntary written informed consent before any study related procedure is performed | X | XX |
| | | 18-70 years of age, inclusive | | |
| | | (continued) | X | XX |
| | Exclusion | Any exclusion criterion | X | Xx |
| | | Inability to swallow tablets | X | Xx |
| | | Presence of any condition or finding which would jeopardize subject safety, impact study result validity, or diminish the subject's ability to undergo all study procedures and assessments | X | Xx |
| | | (continued) | A | Xx |

**Ineligibility Summary of Screen Failures** (continued) Table 8:

| Subjects with<br>Hepatic<br>Impairment/<br>Non-Hepatically<br>Impaired Controls | Inclusion/<br>Exclusion<br>Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | <b>%</b> b |
|---|---|---|---|---|
| | Eligible but<br>Not Enrolled | Any Reason | x | xx |
| | | Time Commitment | X | xx |
| Non-Hepatically<br>Impaired Controls<br>(continued) | Eligible but<br>Not Enrolled<br>(continued) | Concern of Potential Risks | х | XX |
| | | Number of Procedures/Blood Draws | X | xx |
| | | Unable to Contact Subjects | X | xx |
| | | Other | x | xx |

a More than one criterion may be marked per subject.
 b Denominator for percentages is the total number of screen failures.

#### 14.1.2 Demographic Data by Impairment Group

Table 9: Summary of Categorical Demographic and Baseline Characteristics by Site

| | | Duke<br>(N=X) | ) | Saint l<br>(N=X) | | All Su<br>(N=X) | • |
|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % |
| Sex | Male | x | xx | x | xx | x | xx |
| | Female | x | xx | X | xx | x | xx |
| Ethnicity | Not Hispanic or Latino | x | xx | x | xx | x | xx |
| | Hispanic or Latino | x | xx | x | xx | x | xx |
| | Not Reported | x | xx | X | xx | x | xx |
| | Unknown | x | xx | X | xx | X | xx |
| Race | American Indian or Alaska Native | x | xx | x | xx | x | xx |
| | Asian | x | xx | x | xx | x | xx |
| | Native Hawaiian or Other Pacific Islander | X | xx | x | xx | х | xx |
| | Black or African American | x | xx | x | xx | x | xx |
| | White | x | xx | x | xx | x | xx |
| | Multi-Racial | x | xx | x | xx | x | xx |
| | Unknown | x | xx | x | xx | x | xx |

Note: N= All Enrolled Subjects

Table 10: Summary of Continuous Demographic and Baseline Characteristics by Site

| Variable | Statistic | Duke<br>(N=X) | Saint Louis (N=X) | All Subjects (N=X) |
|---|---|---|---|---|
| Age (years) | Mean | xx | xx | xx |
| | Standard Deviation | xx | xx | xx |
| | Median | x | x | x |
| | 25 <sup>th</sup> Quartile | x | x | х |
| | 75 <sup>th</sup> Quartile | x | x | х |
| | Minimum | x | х | х |
| | Maximum | x | X | X |
| Weight* (kg) | Mean | xx | xx | xx |
| | Standard Deviation | xx | XX | xx |
| | Median | x | х | х |
| | 25 <sup>th</sup> Quartile | x | X | X |
| | 75 <sup>th</sup> Quartile | x | X | х |
| | Minimum | x | X | х |
| | Maximum | x | х | х |
| Height (cm) | Mean | xx | xx | xx |
| | Standard Deviation | xx | xx | xx |
| | Median | x | X | x |
| | 25 <sup>th</sup> Quartile | x | X | x |
| | 75 <sup>th</sup> Quartile | x | X | x |
| | Minimum | x | X | x |
| | Maximum | x | X | x |
| BMI (kg/m²) | Mean | xx | xx | xx |
| | Standard Deviation | xx | xx | xx |
| | Median | x | X | x |
| | 25th Quartile | x | X | x |
| | 75th Quartile | x | X | x |
| | Minimum | x | X | x |
| | Maximum | x | X | х |

Note: N=All Enrolled Subjects
\*Weight measured at screening

Table 11: Summary of Categorical Demographic and Baseline Characteristics by Impairment Group

| | | | Mild Hepatic<br>Impairment<br>(N=X) | | Moderate<br>Hepatic<br>Impairment<br>(N=X) | | Severe<br>Hepatic<br>Impairment<br>(N=X) | | Matched<br>Controls<br>(N=X) | | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | X | XX | x | xx | x | xx | x | xx | x | xx |
| | Female | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | X | xx | x | xx | X | xx | x | xx | x | xx |
| | Hispanic or Latino | | | | | | | | | | |
| | Not Reported | | | | | | | | | | |
| | Unknown | ;<br> | | | | | | | | | |
| Race | American Indian or Alaska<br>Native | X | xx | X | XX | x | xx | x | xx | X | xx |
| | Asian | ;<br> | | | | | | | | | |
| | Native Hawaiian or Other<br>Pacific Islander | | | | | | | | | | |
| | Black or African American | | | | | | | | | | |
| | White | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | |
| | Unknown | | | | | | | | | | |

Note: N= All Enrolled Subjects

**Table 12: Summary of Continuous Demographic and Baseline Characteristics by Impairment** Group

| Variable | Statistic | Mild Hepatic<br>Impairment<br>(N=X) | Moderate Hepatic<br>Impairment<br>(N=X) | Severe Hepatic<br>Impairment<br>(N=X) | Matched<br>Controls<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|
| Age (years) | Mean | XX | xx | XX | XX | xx |
| | Standard Deviation | xx | xx | xx | XX | xx |
| | Median | X | x | x | X | x |
| | 25 <sup>th</sup> Quartile | X | x | x | X | x |
| | 75 <sup>th</sup> Quartile | X | x | x | X | x |
| | Minimum | X | x | x | X | x |
| | Maximum | Х | X | x | Х | X |
| Weight* (kg) | Mean | XX | xx | XX | XX | xx |
| | Standard Deviation | XX | xx | xx | XX | xx |
| | Median | Х | X | x | Х | X |
| | 25 <sup>th</sup> Quartile | Х | X | х | X | x |
| | 75 <sup>th</sup> Quartile | Х | X | х | X | x |
| | Minimum | Х | X | х | X | x |
| | Maximum | Х | X | х | X | x |
| Height (cm) | Mean | XX | xx | xx | XX | xx |
| | Standard Deviation | xx | xx | xx | XX | xx |
| | Median | X | X | x | Х | X |
| | 25 <sup>th</sup> Quartile | Х | x | x | Х | x |
| | 75 <sup>th</sup> Quartile | X | X | x | Х | X |
| | Minimum | Х | x | x | Х | x |
| | Maximum | x | X | x | Х | X |
| BMI (kg/m²) | Mean | XX | xx | xx | XX | xx |
| | Standard Deviation | XX | xx | xx | XX | xx |
| | Median | X | х | x | X | x |
| | 25th Quartile | Х | x | x | Х | x |
| | 75th Quartile | X | x | x | X | x |
| | Minimum | X | x | x | X | x |
| | Maximum | X | x | x | X | X |

Note: N=All Enrolled Subjects

#### 14.1.3 Prior and Concurrent Medical Conditions

Table 13: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Impairment Group

| | Impairment | | | | Severe Hepatic<br>Impairment (N=X) | Matched Controls (N=X) | All Subjects (N=X) | S |
|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | | | n | % |
| Any SOC | X | xx | x | xx | | | x | xx |
| [SOC 1] | | | | | | | | |
| [SOC 2] | | | | | | | | |

Note: N= Number of subjects in the Safety Population

n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

## 14.2 Efficacy/Immunogenicity Data

Not Applicable.

#### 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

**Table 14:** Overall Summary of Adverse Events

| | Mild Hepatic<br>Impairment<br>(N=X) | | Moderate Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment<br>(N=X) | | Matched<br>Controls<br>(N=X) | | All Subjects (N = X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % |
| At least one unsolicited adverse event | х | X | х | x | Х | х | Х | X | x | х |
| At least one clinical safety laboratory of mild or greater severity through Day 12 | | x | x | x | х | х | x | x | x | Х |
| At least one related unsolicited adverse event | | X | X | X | x | X | X | x | x | x |
| Mild (Grade 1) | x | x | x | x | х | x | x | X | x | X |
| Moderate (Grade 2) | x | x | x | x | х | x | X | X | X | X |
| Severe (Grade 3) | x | x | x | x | х | x | X | X | X | X |
| Not yet assessed | X | X | X | Х | х | X | X | x | x | X |
| At least one severe (Grade 3) unsolicited adverse event | | X | X | X | X | X | X | X | X | x |
| Related | x | x | x | x | х | X | X | X | X | X |
| Unrelated | X | х | X | х | х | X | Х | X | х | х |

Table 14: **Overall Summary of Adverse Events** (continued)

| | Mild Hepatic<br>Impairment<br>(N=X) | | Moderate Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment<br>(N=X) | | Matched<br>Controls<br>(N=X) | | All Subjects (N = X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % |
| At least one serious adverse event <sup>b</sup> | | x | x | x | X | X | X | X | X | X |
| At least one related, serious adverse event | | х | х | x | X | x | X | X | X | x |
| At least one adverse event leading to early termination <sup>c</sup> | | X | X | x | X | X | X | X | X | X |

 $<sup>\</sup>overline{N = Number of subjects in the Safety Population}$ 

<sup>&</sup>lt;sup>a</sup> Subjects are counted once for each category regardless of the number of events.
<sup>b</sup> A listing of Serious Adverse Events is included in Table 18.

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF.
#### 14.3.1.1 Solicited Adverse Events

Not Applicable.

#### 14.3.1.2 Unsolicited Adverse Events

Table 15: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group – Mild Hepatic Impairment

| MedDRA<br>System Organ | MedDRA<br>Preferred | Day 1-5<br>(N=X) | | | | Day 6-1:<br>(N=X) | 2 | | | Any Tim<br>(N=X) | e Post Dose | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class | Term | n | % | 95% CI | Events | n | % | 95% CI | Events | n | % | 95% CI | Events |
| | Any PT | x | xx | xx, xx | X | x | xx | xx, xx | X | x | XX | xx, xx | х |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |

Note: N = number of subjects in the Safety Population. This table presents number and percentage of subjects. A subject is only counted once per PT/time point.

#### Tables with similar format:

- Table 16: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group Moderate Hepatic Impairment
- Table 17: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group Severe Hepatic Impairment
- Table 18: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Impairment Group Matched Controls

Table 19: Incidence of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Impairment Group

| MedDRA | | | Mild<br>(N = | | tic Im | pairme | ent | | | derate : | Hepat | ic Imp | airme | ent | Seve<br>(N = | ere Hep | oatic I | npairı | nent | | Mat<br>(N = | ched C<br>X) | ontro | ls | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ<br>Class | Preferred<br>Term | Severity | Rela | ted | Not<br>Rela | ted | Tot | tal | Rel | ated | Not<br>Rela | ited | Tot | tal | Rela | ited | Not<br>Rela | ted | Tot | tal | Rela | ted | Not<br>Rela | ted | То | tal |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | Any<br>Severity | X | xx | X | xx | х | xx | X | xx | X | XX | х | xx | X | XX | X | xx | х | xx | X | xx | X | xx | X | xx |
| | | Mild | х | XX | х | xx | X | XX | Х | xx | х | xx | х | xx | X | xx | X | xx | х | xx | х | xx | х | xx | х | xx |
| | | Moderate | x | xx | x | XX | х | xx | х | xx | х | xx | х | XX | х | xx | X | xx | х | XX | x | XX | х | xx | х | xx |
| | | Severe | x | xx | x | XX | х | xx | х | xx | х | xx | х | XX | х | xx | X | xx | х | XX | x | XX | х | xx | х | xx |
| SOC 1 | PT 1 | Any<br>Severity | X | xx | X | xx | х | xx | X | xx | X | XX | х | xx | X | XX | X | xx | х | xx | X | xx | X | xx | X | xx |
| | | Mild | х | xx | х | XX | х | xx | Х | xx | Х | xx | х | XX | х | xx | X | xx | х | XX | x | XX | х | xx | х | xx |
| | | Moderate | х | XX | х | XX | х | xx | Х | xx | Х | xx | х | XX | х | xx | X | xx | х | XX | х | XX | х | xx | х | xx |
| | | Severe | х | XX | х | xx | X | XX | Х | xx | х | xx | х | xx | X | xx | X | xx | х | xx | х | xx | х | xx | х | xx |
| | PT 2 | Any<br>Severity | X | xx | X | xx | х | xx | X | xx | X | XX | х | xx | X | XX | X | xx | х | xx | X | xx | X | xx | X | xx |
| | | Mild | х | XX | х | xx | X | XX | Х | xx | х | xx | х | xx | X | xx | х | xx | х | xx | х | xx | х | xx | х | xx |
| | | Moderate | х | xx | х | XX | х | xx | х | xx | х | XX | х | XX | Х | xx | X | XX | х | XX | X | XX | X | XX | х | xx |
| | | Severe | х | XX | х | xx | X | XX | Х | xx | х | xx | х | xx | X | xx | х | xx | х | xx | х | xx | х | xx | х | xx |

Note: N = Number of subjects in the Safety Population.

# 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

 Table 20:
 Listing of Serious Adverse Events

| Adverse<br>Event | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term | No. of Days Post<br>Dose | Duration | No. of<br>Days<br>Post<br>Dose the<br>Event<br>Became<br>Serious | Reason<br>Reported<br>as an<br>SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Impairme | nt Group: Su | bject ID: | AE Number: | | | | | | | | | |
| Comments | : | | | | | | | | | | | |
| Impairme | nt Group: Su | bject ID: | AE Number: | | | | | | | | | |
| Comments | : | | | | | | | | | | | |

| Adverse<br>Event | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term | No. of Days<br>Post Dose | Duration | No. of Days Post Dose the Event Became Serious | Reason<br>Reported<br>as an<br>SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Impairm | ent Group: S | Subject ID: | AE Number: | <b>,</b> | | <del>,</del> | | | <del>,</del> | | | |
| Comment | s: | | | | | | | | | | | |
| Impairm | ent Group: S | Subject ID: | AE Number: | | | | | | | | | |
| Comment | s: | | | | | | | | | | | ' |

# 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

# 14.3.4 Abnormal Laboratory Value Listings (by Subject)

### **Table 22:** Listing of Abnormal Laboratory Results - Chemistry

| Impairment Group | Subject<br>ID | Sex | Age (years) | Actual Study<br>Day | Laboratory Parameter (Units) | Result (Severity) |
|---|---|---|---|---|---|---|

| Impairment<br>Group | Subject<br>ID | Sex | Age (years) | Planned Time Point | Actual Study Day | Laboratory Parameter (Units) | Result (Severity) |
|---|---|---|---|---|---|---|---|

| Impairment Group | Subject<br>ID | Sex | Age (years) | Planned Time Point | Actual Study Day | Laboratory Parameter (Units) | Result (Severity) |
|---|---|---|---|---|---|---|---|

**Table 25:** Listing of Abnormal Laboratory Results - Coagulation

| Impairment Group | Subject<br>ID | Sex | Age (years) | Planned Time Point | Actual Study Day | Laboratory Parameter (Units) | Result (Severity) |
|---|---|---|---|---|---|---|---|

# 14.3.5 Displays of Laboratory Results

# 14.3.5.1 Chemistry Results

Table 26: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Chemistry Parameter

| | | | None | | Mild/<br>Grade 1 | 1 | Modera<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | x | xx | х | xx | х | xx | х | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 26: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Chemistry Parameter (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | 1 | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

### Tables with similar format:

Table 27: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Total Bilirubin

Table 28: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Serum Albumin

inpendin it fuels intern eps

Table 29: Chemistry Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – Potassium

| | | | None | | Mild/<br>Grade<br>(Low) | | Mild/<br>Grade<br>(High) | | Moder:<br>Grade<br>(Low) | | Moder<br>Grade<br>(High) | 2 | Severe/<br>Grade<br>(Low) | | Severe/<br>Grade (High) | | Missing | 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic<br>Impairment | X | X | XX | X | XX | Х | xx | X | xx | Х | xx | X | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

| | | | None | | Mild/<br>Grade<br>(Low) | 1 | Mild/<br>Grade<br>(High) | 1 | Modera<br>Grade 2<br>(Low) | | Modera<br>Grade 2<br>(High) | | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | | Missing | , |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Day 12 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Max Severity Post<br>Baseline | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table 30: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Magnesium

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | X | xx | x | xx | X | xx | X | xx | x | XX |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 30: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Magnesium (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % n | | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Appendix 1: Table Mock-Ups

Table 31: Chemistry Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – Calcium

| | | | None | | Mild/<br>Grade<br>(Low) | e 1 | Mild/<br>Grade<br>(High) | | Moder<br>Grade<br>(Low) | | Moder<br>Grade<br>(High) | 2 | Severe/<br>Grade<br>(Low) | | Severe/<br>Grade<br>(High) | | Missing | · |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic<br>Impairment | x | X | XX | X | XX | X | xx | X | xx | X | XX | X | xx | x | xx | X | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table 31: Chemistry Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – Calcium (continued)

| | | | None | | Mild/<br>Grade<br>(Low) | 1 | Mild/<br>Grade<br>(High) | 1 | Modera<br>Grade 2<br>(Low) | | Modera<br>Grade 2<br>(High) | | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | | Missing | , |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Day 12 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Max Severity Post<br>Baseline | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table with similar format:

Table 32: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Serum Creatinine

Table 33: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – BUN

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | x | XX | x | xx | X | xx | x | xx | X | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 33: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – BUN (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | ′ | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | n % n | | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

### Tables with Similar format:

Table 34: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Alkaline Phosphatase

Table 35: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – ALT

Table 36: Chemistry Laboratory Results by Maximum Severity, Time Point, and Impairment Group – AST

Table 37: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Any Chemistry Parameter

| | | | Mild/<br>Grade 1 | | Modera<br>Grade 2 | | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | X | xx | X | xx | X | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N= Number of subjects in the Safety Population with labs available at each visit.

### Tables with similar format:

- Table 38: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Total Bilirubin
- Table 39: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Serum Albumin

Table 40: Abnormal Chemistry Laboratory Results Related to Study Treatment by Range, Maximum Severity, Time Point, and Impairment Group – Potassium

| | | | Mild/<br>Grade 1<br>(Low) | I | Mild/<br>Grade 1<br>(High) | Į. | Moderate<br>Grade 2<br>(Low) | e/ | Moderat<br>Grade 2<br>(High) | e/ | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | x | xx | x | xx | X | xx | x | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

| | | | Mild/<br>Grade 1<br>(Low) | | Mild/<br>Grade 1<br>(High) | | Moderate<br>Grade 2<br>(Low) | <u>e</u> / | Moderate<br>Grade 2<br>(High) | e/ | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

Table 41: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Magnesium

| | | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | e/ | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | x | xx | X | xx | X | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |

Table 42: Abnormal Chemistry Laboratory Results Related to Study Treatment by Range, Maximum Severity, Time Point, and Impairment Group – Calcium

| | | | Mild/<br>Grade 1<br>(Low) | I | Mild/<br>Grade 1<br>(High) | Į. | Moderate<br>Grade 2<br>(Low) | e/ | Moderat<br>Grade 2<br>(High) | e/ | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | x | xx | x | xx | X | xx | x | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

Table 42: Abnormal Chemistry Laboratory Results Related to Study Treatment by Range, Maximum Severity, Time Point, and Impairment Group – Calcium (continued)

| | | | Mild/<br>Grade 1<br>(Low) | | Mild/<br>Grade 1<br>(High) | | Moderate<br>Grade 2<br>(Low) | ·/ | Moderate<br>Grade 2<br>(High) | <u>*</u> / | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

Table with Similar Format:

Table 43: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Serum Creatinine

Table 44: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – BUN

| | | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | e/ | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | х | Х | XX | X | xx | X | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |

### Tables with Similar Format:

- Table 45: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Alkaline Phosphatase
- Table 46: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group ALT
- Table 47: Abnormal Chemistry Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group AST

Table 48: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group – Total Bilirubin (mg/dL)

| ax |
|-----|
| I.X |

Table 48: Chemistry Laboratory Statistics by Time Point, and Impairment Group – Total Bilirubin (mg/dL) (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 12, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Note: N= Number of subjects in the Safety Population with labs available at each visit.

#### Tables with similar format:

| Table 49: | Chemistry Labora | tory Summary | Statistics by | Time Point and Im | pairment Groui | o – Serum Albumin (g/dL) |
|---|---|---|---|---|---|---|

- Table 50: Chemistry Laboratory Summary Statistics by Range, Time Point, and Impairment Group Potassium (mmol/dL)
- Table 51: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group Magnesium (mg/dL)
- Table 52: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group Calcium (mg/dL)
- Table 53: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group Serum Creatinine (mg/dL)
- Table 54: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group BUN (mg/dL)
- Table 55: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group Alkaline Phosphatase (U/L)
- Table 56: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group ALT (U/L)
- Table 57: Chemistry Laboratory Summary Statistics by Time Point and Impairment Group AST (U/L)

## 14.3.5.2 Hematology Results

Table 58: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Hematology Parameter

| | | | None | | Mild/<br>Grade 1 | | | Moderate/<br>Grade 2 | | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | x | xx | x | xx | x | xx | х | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 58: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Hematology Parameter (continued)

| | | | | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

### Tables with similar format:

Table 59: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Hematocrit

Table 60: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Hemoglobin

Table 61: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Red Blood Cell Count

Table 62: Hematology Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – White Blood Cell Count

| | | | None | | Mild/<br>Grade<br>(Low) | 1 | Mild/<br>Grade<br>(High) | | Moder:<br>Grade<br>(Low) | | Moder<br>Grade<br>(High) | 2 | Severe/<br>Grade (Low) | | Severe/<br>Grade<br>(High) | | Missing | 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic<br>Impairment | X | Х | xx | X | xx | х | xx | Х | xx | X | xx | x | xx | x | xx | X | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table 62: Hematology Laboratory Results by Range, Maximum Severity, Time Point, and Impairment Group – White Blood Cell Count (continued)

| | | | None | | Mild/<br>Grade (Low) | 1 | Mild/<br>Grade (High) | 1 | Modera<br>Grade 2<br>(Low) | | Modera<br>Grade 2<br>(High) | | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | | Missing | Į. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Day 12 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Max Severity Post<br>Baseline | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table 63: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Neutrophils

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | x | xx | x | xx | х | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Appendix 1: Table Mock-Ups

Table 63: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Neutrophils (continued)

| | | | | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

### Tables with similar format

Table 64: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Eosinophils

Table 65: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Basophils

Table 66: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Lymphocytes

Table 67: Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Absolute Monocytes

**Table 68:** Hematology Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Platelets

Table 69: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Any Hematology Parameter

| | | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | X | XX | X | XX | x | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
### Tables with similar format:

- Table 70: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Hematocrit
- Table 71: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Hemoglobin
- Table 72: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Red Blood Cell Count

Table 73: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – White Blood Cell Count

| | | | Mild/<br>Grade 1<br>(Low) | | Mild/<br>Grade 1<br>(High) | | Moderate<br>Grade 2<br>(Low) | e/ | Moderate/<br>Grade 2<br>(High) | | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | x | xx | x | xx | x | xx | x | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

Table 73: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – White Blood Cell Count (continued)

| | | | Grade 1 | | Grade 1 | | Grade 2 | | Moderate/<br>Grade 2<br>(High) | | Severe/<br>Grade 3<br>(Low) | | Severe/<br>Grade 3<br>(High) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N=Number of subjects in the Safety Population with labs available at each visit.

Table 74: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Absolute Neutrophils

| | | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | e/ | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | Х | x | xx | x | XX | Х | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

### Tables with similar format

- Table 75: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Absolute Eosinophils
- Table 76: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Absolute Basophils
- Table 77: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Absolute Lymphocytes
- Table 78: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Absolute Monocytes
- Table 79: Abnormal Hematology Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Platelets

Table 80: Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Hematocrit (%)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Mild Hepatic Impairment | x | xx.x | xx.x | xx.x | xx.x, xx.x |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 2, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 80: Hematology Laboratory Statistics by Time Point and Impairment Group – Hematocrit (%) (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 12, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Note: N= Number of subjects in the Safety Population with labs available at each visit.

## Tables with similar format:

| Table 81: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Hemoglobin (g/dL) |
|---|---|
| Table 82: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Red Blood Cell Count (x1012/L) |
| Table 83: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – White Blood Cell Count (x109/L) |
| Table 84: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Neutrophils (x109/L) |
| Table 85: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Eosinophils (x109/L) |
| Table 86: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Basophils (x109/L) |
| <b>Table 87:</b> | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Lymphocytes (x109/L) |
| Table 88: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Absolute Monocytes (x109/L) |
| Table 89: | Hematology Laboratory Summary Statistics by Time Point and Impairment Group – Platelets (x109/L) |

#### 14.3.5.3 **Urinalysis Results**

Table 90: Urinalysis Laboratory Results by Parameter, Time Point, and Impairment Group

| | | | Urine Bloo | d | Urine Prote | ein | Urine Glucose | | Any Param | ieter |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | х | xx | x | xx | x | xx | x | xx |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |

N= Number in the safety population with labs available at each visit. n= Number with positive dipstick results.

Table 91: Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Urinalysis Parameter

| | | None | | Mild/<br>Grade | 1 | Moderat<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | x | xx | х | xx | х | xx | X | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 91: Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Any Urinalysis Parameter (continued)

| | | | | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

### Tables with similar format:

Table 92: Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Protein

Table 93: Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Glucose

Table 94: Urinalysis Laboratory Results by Maximum Severity, Time Point, and Impairment Group – Urine Blood

Table 95: Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – Any Urinalysis Parameter

| | | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | e/ | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | Х | x | xx | x | XX | Х | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

### Tables with similar format:

- Table 96: Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Protein
- Table 97: Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Glucose
- Table 98: Abnormal Urinalysis Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group Urine Blood

# Table 99: Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Blood (rbc/hpf)

[Implementation Note: Microscopic urine analysis is only performed if there is an abnormal urine result. Therefore, there may not be enough data to present this table.]

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Mild Hepatic Impairment | X | xx.x | xx.x | xx.x | xx.x, xx.x |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 2, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 99: Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Blood (rbc/hpf) (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 12 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Note: N= Number of subjects in the Safety Population with a positive urine dipstick result and with labs available at each visit.

# Table 100: Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Protein

[Implementation Note: Microscopic urine analysis is only performed if there is an abnormal urine result. Therefore, there may not be enough data to present this table.]

| | | | Negative | ! | Trace | | 1+ | | 2+ | | 3+ | | 4+ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | X | xx | x | xx | X | xx | x | XX | X | xx | X | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

#### 

| | | | Negativ | e | Trace | | 1+ | | 2+ | | 3+ | | 4+ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |
| Max Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

### Table with similar format:

Table 101: Urinalysis Laboratory Summary Statistics by Time Point and Impairment Group – Glucose

## 14.3.5.4 Coagulation Results

Table 102: Coagulation Laboratory Results by Maximum Severity, Time Point, and Impairment Group – INR

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | X | x | xx | X | xx | х | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Appendix 1: Table Mock-Ups

Table 102: Coagulation Laboratory Results by Maximum Severity, Time Point, and Impairment Group – INR (continued)

| | | | None | | | Mild/<br>Grade 1 | | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

Table 103: Abnormal Coagulation Laboratory Results Related to Study Treatment by Maximum Severity, Time Point, and Impairment Group – INR

| | | | Mild/<br>Grade 1 | | Moderat<br>Grade 2 | <b>e</b> / | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % |
| Baseline | Mild Hepatic Impairment | x | x | xx | х | xx | X | XX |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | |
| | Matched Controls | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population with labs available at each visit.

Table 104: Coagulation Laboratory Summary Statistics by Time Point and Impairment Group – INR

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Mild Hepatic Impairment | x | xx.x | XX.X | xx.x | xx.x, xx.x |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 2 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 2, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 104: Coagulation Laboratory Summary Statistics by Time Point and Impairment Group – INR (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 12, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Note: N= Number of subjects in the Safety Population with labs available at each visit.

Appendix 1: Table Mock-Ups

Table 105: Chemistry Shift Tables by Time Point and Impairment Group – Total Bilirubin

[Implementation Note: If there is no low range then those columns will be removed.]

| | Mild H<br>(N=X)<br>Baselin | epatic Impa<br>e | irment | | (N=X)<br>Baseline | | | | Severe Hepatic Impairment (N=X) Baseline | | | | Matched Controls (N=X) Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day Post Dose | Low | Normal | High | Total | Low | Normal | High | Total | Low | Normal | High | Total | Low | Normal | High | Total |
| Day 2 | | | | | | | | | | | | | | | | |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 5 | | | | | | | | | | | | | | | | |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 12 | | • | | | | | | • | | | | | | | | |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

## Tables with similar format:

Table 106: Chemistry Shift Tables by Time Point and Impairment Group – Serum Albumin

Table 107: Chemistry Shift Tables by Time Point and Impairment Group – Potassium

Table 108: Chemistry Shift Tables by Time Point and Impairment Group – Magnesium

**Table 128:** 

| <b>Table 109:</b> | Chemistry Shift Tables by Time Point and Impairment Group - Calcium |
|---|---|
| <b>Table 110:</b> | Chemistry Shift Tables by Time Point and Impairment Group – Serum Creatinine |
| <b>Table 111:</b> | Chemistry Shift Tables by Time Point and Impairment Group – BUN |
| <b>Table 112:</b> | Chemistry Shift Tables by Time Point and Impairment Group – Alkaline Phosphatase |
| <b>Table 113:</b> | Chemistry Shift Tables by Time Point and Impairment Group – ALT |
| <b>Table 114:</b> | Chemistry Shift Tables by Time Point and Impairment Group – AST |
| <b>Table 115:</b> | Hematology Shift Tables by Time Point and Impairment Group – Hematocrit |
| <b>Table 116:</b> | Hematology Shift Tables by Time Point and Impairment Group – Hemoglobin |
| <b>Table 117:</b> | Hematology Shift Tables by Time Point and Impairment Group – Red Blood Cell Count |
| <b>Table 118:</b> | Hematology Shift Tables by Time Point and Impairment Group – White Blood Cell Count |
| <b>Table 119:</b> | Hematology Shift Tables by Time Point and Impairment Group – Neutrophils |
| <b>Table 120:</b> | Hematology Shift Tables by Time Point and Impairment Group – Eosinophils |
| <b>Table 121:</b> | Hematology Shift Tables by Time Point and Impairment Group – Basophils |
| <b>Table 122:</b> | Hematology Shift Tables by Time Point and Impairment Group – Lymphocytes |
| <b>Table 123:</b> | Hematology Shift Tables by Time Point and Impairment Group – Monocytes |
| <b>Table 124:</b> | Hematology Shift Tables by Time Point and Impairment Group – Platelets |
| <b>Table 125:</b> | Coagulation Shift Tables by Time Point and Impairment Group – INR |
| <b>Table 126:</b> | Urinalysis Shift Tables by Time Point and Impairment Group – Protein |
| <b>Table 127:</b> | Urinalysis Shift Tables by Time Point and Impairment Group – Glucose |

**Urinalysis Shift Tables by Time Point and Impairment Group – Blood** 

# 14.3.6 Displays of Vital Signs

Table 129: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Any Assessment

| | | | None | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % |
| Admission | Mild Hepatic Impairment | x | X | xx | X | xx | x | xx | x | xx |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Baseline | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 1 hour post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 2 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 4 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |

Table 129: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Any Assessment (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % |
| 5 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 6 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 8 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 12 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 16 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |

Table 129: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Any Assessment (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | 1 | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % |
| 24 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| 36 hours post-dose | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Day 3 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Day 4 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |

Table 129: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Any Assessment (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | |
| | Moderate Hepatic Impairment | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | |
| | Matched Controls | | | | | | | | | |

Table with similar format:

Table 130: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Oral Temperature

Table 131: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Pulse

| | | | None | | Mild<br>(Low) | | Mild<br>(High) | | Moder<br>(Low) | | Moder<br>(High) | | Severe<br>(Low) | | Severe<br>(High) | | Missin | ıg |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Admission | Mild Hepatic<br>Impairment | X | Х | XX | X | XX | X | xx | X | xx | Х | XX | Х | xx | X | xx | X | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Baseline | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 1 hour post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 2 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Appendix 1: Table Mock-Ups

Table 131: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Pulse (continued)

| | | | None | | Mild<br>(Low) | | Mild<br>(High) | ) | Moder<br>(Low) | | Moder<br>(High) | | Severe<br>(Low) | | Severe<br>(High) | | Missin | ıg |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| 4 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 5 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 6 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 8 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Appendix 1: Table Mock-Ups

Table 131: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Pulse (continued)

| | | | None | | Mild<br>(Low) | | Mild<br>(High) | ) | Moder<br>(Low) | | Moder<br>(High) | | Severe<br>(Low) | | Severe<br>(High) | | Missin | ıg |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| 12 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 16 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 24 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| 36 hours post-dose | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table 131: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Pulse (continued)

| | | | None | | Mild<br>(Low) | | Mild<br>(High) | ) | Moder<br>(Low) | | Moder<br>(High) | | Severe<br>(Low) | | Severe<br>(High) | | Missin | ıg |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Day 3 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 4 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 5 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |
| Day 12 | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Table 131: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Pulse (continued)

| | | | None | | Mild<br>(Low) | | Mild<br>(High) | | Modera<br>(Low) | ite | Modera<br>(High) | ite | Severe<br>(Low) | | Severe<br>(High) | | Missing | 5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | Mild Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Severe Hepatic<br>Impairment | | | | | | | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N = [define the population for this table, e.g., Number of subjects in the Safety Population]

Table with similar format:

Table 132: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Systolic Blood Pressure

Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diastolic Blood Pressure

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | e/ | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Admission | Mild Hepatic Impairment | X | x | xx | x | xx | x | xx | x | xx | x | xx |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 1 hour post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 2 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 4 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diastolic Blood Pressure (continued)

| | | | None | | Mild/<br>Grade | 1 | Moder<br>Grade | | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| 5 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 6 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 8 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 12 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 16 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diastolic Blood Pressure (continued)

| | | | None | | Mild/<br>Grade | 1 | Moder<br>Grade | | Severe/<br>Grade 3 | | Missin | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| 24 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| 36 hours post-dose | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 3 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 4 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Table 133: Vital Signs by Maximum Severity, Time Point, and Impairment Group – Diastolic Blood Pressure (continued)

| | | | None | | Mild/<br>Grade 1 | | Moderate<br>Grade 2 | / | Severe/<br>Grade 3 | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Impairment Group | N | n | % | n | % | n | % | n | % | n | % |
| Day 12 | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | | | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | | | | | | | |
| | Severe Hepatic Impairment | | | | | | | | | | | |
| | Matched Controls | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population at each visit.
Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral Temperature

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Admission | Mild Hepatic Impairment | x | xx.x | XX.X | xx.x | xx.x, xx.x |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 1 hour post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 1 hour post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 2 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 2 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral Temperature (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| 4 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 4 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 5 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 5 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 6 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 6 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral Temperature (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| 8 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 8 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 12 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 12 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 16 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 16 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral Temperature (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| 24 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 24 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 36 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 36 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 3 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 3, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral Temperature (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 4 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 4, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Appendix 1: Table Mock-Ups

Table 134: Vital Signs Summary Statistics by Time Point and Impairment Group – Oral Temperature (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Note: N= Number of subjects in the Safety Population at ea | Note: N= Number of subjects in the Safety Population at each visit | | | | | |

#### Tables with similar format:

Table 135: Vital Signs Summary Statistics by Time Point and Impairment Group – Pulse

Table 136: Vital Signs Summary Statistics by Time Point and Impairment Group – Systolic Blood Pressure

Table 137: Vital Signs Summary Statistics by Time Point and Impairment Group – Diastolic Blood Pressure

Table 138: Summary of Abnormal Physical Exam Findings by Impairment Group

| Time Point | | Mild H<br>Impair<br>(N=X) | Mild Hepatic<br>Impairment<br>(N=X) | | Moderate Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment (N=X) | | Matched Controls (N=X) | | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Time I ome | Body System | n | % | n | % | n | % | n | % | n | % |
| Admission | Any Body System | x | xx | x | xx | X | XX | x | xx | x | XX |
| | Abdomen | | | | | | | | | | |
| | Cardiovascular/Heart | | | | | | | | | | |
| | Extremities | | | | | | | | | | |
| | General Appearance | | | | | | | | | | |
| | HEENT | | | | | | | | | | |
| | Lymph Nodes | | | | | | | | | | |
| | Musculoskeletal | | | | | | | | | | |
| | Neck (Thyroid) | | | | | | | | | | |
| | Neurological | | | | | | | | | | |
| | Pulmonary/Chest | | | | | | | | | | |
| | Skin | | | | | | | | | | |
| Day 12 | Any Body System | x | xx | x | xx | x | XX | x | xx | x | xx |
| | Abdomen | | | | | | | | | | |
| | Cardiovascular/Heart | | | | | | | | | | |
| | Extremities | | | | | | | | | | |
| | General Appearance | | | | | | | | | | |
| | HEENT | | | | | | | | | | |
| | Lymph Nodes | | | | | | | | | | |

Appendix 1: Table Mock-Ups

Table 138: Summary of Abnormal Physical Exam Findings by Impairment Group (continued)

| Time Point | | Impairment | | Moderate Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment (N=X) | | Matched Controls (N=X) | | All Subjection (N=X) | ets |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Tome | Body System | n | % | n | % | n | % | n | % | n | % |
| | Musculoskeletal | | | | | | | | | | |
| | Neck (Thyroid) | | | | | | | | | | |
| | Neurological | | | | | | | | | | |
| | Pulmonary/Chest | | | | | | | | | | |
| | Skin | | | | | | | | | | |

Note: N= Number of subjects in the Safety Population at each visit

n = Number of subjects with physical exam findings.

Table 139: Physical Exam Summary Statistics by Time Point and Impairment Group – Weight

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Admission | Mild Hepatic Impairment | x | xx.x | xx.x | xx.x | xx.x, xx.x |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 1 hour post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 1 hour post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 2 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 2 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 139: Physical Exam Summary Statistics by Time Point and Impairment Group – Weight (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| 4 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 4 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 5 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 5 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 6 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 6 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 139: Physical Exam Summary Statistics by Time Point and Impairment Group – Weight (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| 8 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 8 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 12 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 12 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 16 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 16 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 139: Physical Exam Summary Statistics by Time Point and Impairment Group – Weight (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| 24 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 24 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 36 hours post-dose | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| 36 hours post-dose, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 3 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 3, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Table 139: Physical Exam Summary Statistics by Time Point and Impairment Group – Weight (continued)

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 4 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 4, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 5, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12, Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

| Time Point | Impairment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Max Severity Post Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |

Note: N= Number of subjects in the Safety Population at each visit

Statistical Analysis Plan - DMID Protocol: 13-0053 Version 2.0 Appendix 1: Table Mock-Ups 08 May 2024

## 14.4 Summary of Concomitant Medications

Table 140: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Impairment Group

| WHO Drug Code<br>Level 1, Anatomic | WHO Drug Code<br>Level 2,<br>Therapeutic | Mild Hepatic<br>Impairment<br>(N=X) | | Moderate<br>Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment<br>(N=X) | | Matched<br>Controls (N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Subgroup | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | x | xx | X | xx | | | | | X | xx |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |

N = Number of subjects in the Safety Population

n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

Statistical Analysis Plan - DMID Protocol: 13-0053 Version 2.0 Appendix 1: Table Mock-Ups 08 May 2024

#### 14.5 Other Safety Measures

Table 141: ECG Summary Statistics by Time Point and Impairment Group – RR

| Time Point | Impairment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Admission | Mild Hepatic Impairment | Х | xx.x | XX.X | xx.x | xx.x, xx.x |
| | Moderate Hepatic<br>Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Day 12 | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Change from Baseline | Mild Hepatic Impairment | | | | | |
| | Moderate Hepatic<br>Impairment | | | | | |
| | Severe Hepatic Impairment | | | | | |
| | Matched Controls | | | | | |
| Note: N= Number of subjects | in the Safety Population at each visit | t. | | • | | • |

#### Tables with similar format:

Table 142: ECG Summary Statistics by Time Point and Impairment Group – QRS

Table 143: ECG Summary Statistics by Time Point and Impairment Group – QT

Table 144: ECG Summary Statistics by Time Point and Impairment Group – QTcF

Table 145: ECG Summary Statistics by Time Point and Impairment Group – PR

Table 146: ECG Summary Statistics by Time Point and Impairment Group – Ventricular Rate

Statistical Analysis Plan - DMID Protocol: 13-0053 Version 2.0 Appendix 1: Table Mock-Ups 08 May 2024

Table 147: Number and Percentage of Subjects Experiencing ECG Events by Symptom, and Impairment Group

| | | Mild Hepatic<br>Impairment<br>(N=X) | | Imp | Moderate Hepatic<br>Impairment<br>(N=X) | | Severe Hepatic<br>Impairment<br>(N=X) | | | Matched Controls<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Visit | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | Admission | x | xx | x.x, x.x | х | xx | x.x, x.x | х | xx | x.x, x.x | X | xx | x.x, x.x |
| | Day 12 | | | | | | | | | | | | |
| Bradycardia | Admission | | | | | | | | | | | | |
| | Day 12 | | | | | | | | | | | | |
| Tachycardia | Admission | | | | | | | | | | | | |
| | Day 12 | | | | | | | | | | | | |
| Conduction System<br>Disease | Admission | | | | | | | | | | | | |
| | Day 12 | | | | | | | | | | | | |
| Arrhythmia | Admission | | | | | | | | | | | | |
| | Day 12 | | | | | | | | | | | | |
| Brugada Pattern | Admission | | | | | | | | | | | | |
| | Day 12 | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population at each visit.

#### 14.6 Pharmacokinetics Results

Table 148: Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours)

– Mild Hepatic Impairment

| | Pre-<br>Dose | 1 | 2 | 4 | 5 | 6 | 8 | 12 | 16 | 24 | 36 | 48 | 72 | 96 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 001 | | | | | | | | | | | | | | |
| 002 | | | | | | | | | | | | | | |
| 003 | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | |
| N Not Evaluable | | | | | | | | | | | | | | |
| Number < LLOQ <sup>a</sup> | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> LLOQ=10 ng/mL

Tables with similar format:

Table 149: Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours)

– Moderate Hepatic Impairment

Table 150: Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours)

– Severe Hepatic Impairment

Table 151: Individual and Summary Statistics for Plasma Concentrations by Nominal Time (hours)

- Matched Controls

Statistical Analysis Plan - DMID Protocol: 13-0053

Appendix 1: Table Mock-Ups

Version 2.0

08 May 2024

Table 152: Individual and Summary Statistics for Noncompartmental PK Parameters – Mild Hepatic Impairment

| Subject ID | AUC0-last<br>(ng·hr/mL) | AUC₀-∞<br>(ng·hr/mL) | T <sub>max (hr)</sub> | Cmax<br>(ng/mL) | CL/F<br>(L/hr) | V <sub>d</sub> /F | t <sub>1/2)</sub> (hr) |
|---|---|---|---|---|---|---|---|
| 001 | | | | | | | |
| 002 | | | | | | | |
| 003 | | | | | | | |
| N | | | | | | | |
| Mean | | | | | | | |
| SD | | | | | | | |
| Min | | | | | | | |
| Max | | | | | | | |
| CV % | | | | | | | |
| GM | | | | | | | |

Tables with similar format:

- Table 153: Individual and Summary Statistics for Noncompartmental PK Parameters Moderate Hepatic Impairment
- Table 154: Individual and Summary Statistics for Noncompartmental PK Parameters Severe Hepatic Impairment
- Table 155: Individual and Summary Statistics for Noncompartmental PK Parameters Matched Controls

### **Table 156:** Estimated Impairment Group Fold Change for Noncompartmental PK Parameters

[Implementation Note: The site column will only be included if the group by site interaction is significant at a p-value < 0.10 level.]

| Site | Impairment Group | Statistic | AUC <sub>0-last</sub> (ng·hr/mL) | AUC <sub>0-∞</sub> (ng·hr/mL) | C <sub>max</sub><br>(ng/mL) |
|---|---|---|---|---|---|
| Duke | Mild | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Moderate | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Severe | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Matched Controls | Mean | | | |
| | | 90% CI of Mean | | | |
| Saint Louis | Mild | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Moderate | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Severe | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Matched Controls | Mean | | | |
| | | 90% CI of Mean | | | |
| Overall | Mild | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |

**Table 156:** Estimated Impairment Group Fold Change for Noncompartmental PK Parameters *(continued)* 

| Site | Impairment Group | Statistic | AUC <sub>0-last</sub> (ng·hr/mL) | AUC₀-∞<br>(ng·hr/mL) | C <sub>max</sub> (ng/mL) |
|---|---|---|---|---|---|
| | | 90% CI of Mean | | | |
| | Moderate | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Severe | Mean | | | |
| | | 90% CI of Mean | | | |
| | | Fold Change <sup>a</sup> | | | |
| | | 90% CI of Mean | | | |
| | Matched Controls | Mean | | | |
| | | 90% CI of Mean | | | |

<sup>&</sup>lt;sup>a</sup> Comparison is to matched controls

Statistical Analysis Plan - DMID Protocol: 13-0053

Appendix 1: Table Mock-Ups

Version 2.0
08 May 2024

### **Table 157:** Estimated Impairment Group Shift for Noncompartmental PK Parameters

[Implementation Note: Site column will only be included if confidence intervals between sites do not overlap.]

| GA. | | Q | T <sub>max</sub> |
|-------------|------------------|---------------------|------------------|
| Site | Impairment Group | Statistic | (h) |
| Duke | Mild | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Moderate | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Severe | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Matched Controls | Median | |
| | | 90% CI <sup>a</sup> | |
| Saint Louis | Mild | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Moderate | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Severe | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Matched Controls | Median | |
| | | 90% CI <sup>a</sup> | |

Table 157: Estimated Impairment Group Shift for Noncompartmental PK Parameters (continued)

| Site | Impairment Group | Statistic | T <sub>max</sub> |
|---------|------------------|---------------------|------------------|
| Overall | Mild | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Moderate | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Severe | Median | |
| | | 90% CI <sup>a</sup> | |
| | | Shift <sup>b</sup> | |
| | | 90% CI <sup>a</sup> | |
| | Matched Controls | Median | |
| | | 90% CI <sup>a</sup> | |

<sup>&</sup>lt;sup>a</sup> Confidence limits will be estimated using the inverted rank score method.

<sup>&</sup>lt;sup>b</sup> Comparison is to matched controls

# APPENDIX 2. FIGURE MOCK-UPS

## LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram |
|---|---|
| Figure 2: | Schematic of Study Design |
| Figure 3: | Frequency of Related Adverse Events by MedDRA System Organ Class, Severity, and Impairment Group |
| Figure 4: | Incidence of Related Adverse Events by MedDRA® System Organ Class, Maximum Severity, and Impairment Group |
| Figure 5: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – Total Bilirubin |
| Figure 6: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – Serum Albumin |
| Figure 7 | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – Potassium |
| Figure 8: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – Magnesium |
| Figure 9: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – Calcium |
| Figure 10: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Serum Creatinine |
| Figure 11: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – BUN |
| Figure 12: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Alkaline Phosphatase |
| Figure 13: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – ALT |
| Figure 14: | Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – AST |
| Figure 15: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Hematocrit |
| Figure 16: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Hemoglobin |
| Figure 17: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Red Blood Cell Count |
| Figure 18: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – White Blood Cell Count |
| Figure 19: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – Neutrophils |

# LIST OF FIGURES (continued)

| Figure 20: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – Eosinophils |
|---|---|
| Figure 21: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – Basophils |
| Figure 22: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – Lymphocytes |
| Figure 23: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – Monocytes |
| Figure 24: | Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – Platelets |
| Figure 25: | Coagulation Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – INR |
| Figure 26: | Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Mild Hepatic Impairment |
| Figure 27 | Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Moderate Hepatic Impairment |
| Figure 28: | Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Severe Hepatic Impairment |
| Figure 29: | Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Matched Controls |
| Figure 30: | Linear Plot of Pretomanid Concentration Profiles by Nominal Time for Subjects with Mild Hepatic Impairment and Their Matched Controls |
| Figure 31: | Linear Plot of Pretomanid Concentration Profiles by Nominal Time for Subjects with Moderate Hepatic Impairment and Their Matched Controls |
| Figure 32: | Linear Plot of Pretomanid Concentration Profiles by Nominal Time for Subjects with Severe Hepatic Impairment and Their Matched Controls |
| Figure 33: | Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time – Mild Hepatic Impairment |
| Figure 34: | Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time – Moderate Hepatic Impairment |
| Figure 35: | Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time – Severe Hepatic Impairment |
| Figure 36: | Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time – Matched Controls |
| Figure 37: | Linear Plots of Mean Pretomanid Plasma Concentration by Nominal Time178 |
| Figure 38: | Semilogarithmic Plots of Mean Pretomanid Plasma Concentration by Nominal Time179 |

# LIST OF FIGURES (continued)

| Figure 39: | $Impairment\ Group\ Summary\ for\ Noncompartmental\ PK\ Parameters-C_{max}180$ |
|---|---|
| Figure 40: | $Impairment\ Group\ Summary\ for\ Noncompartmental\ PK\ Parameters-T_{max}\180$ |
| Figure 41: | Impairment Group Summary for Noncompartmental PK Parameters – $AUC_{(0-\infty)}$ 180 |
| Figure 42: | $Impairment\ Group\ Summary\ for\ Noncompartmental\ PK\ Parameters\ -AUC_{(0\text{-last})}\ 180$ |
| Figure 43: | $Impairment\ Group\ Summary\ for\ Noncompartmental\ PK\ Parameters-CL/F180$ |
| Figure 44: | Impairment Group Summary for Noncompartmental PK Parameters – V <sub>d</sub> /F180 |

#### 10.1 Disposition of Subjects

Figure 1: CONSORT Flow Diagram



Figure 2: Schematic of Study Design



<sup>&</sup>lt;sup>1</sup>Group 4a is referring to the non-hepatically impaired controls matched with Group 1

<sup>&</sup>lt;sup>2</sup>Group 4b is referring to the non-hepatically impaired controls matched with Group 2

<sup>&</sup>lt;sup>3</sup>Group 4c is referring to the non-hepatically impaired controls matched with Group 3

# 14.2.2 Efficacy/Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Not Applicable.

#### 14.3.1.2 Unsolicited Adverse Events

# Figure 3: Frequency of Related Adverse Events by MedDRA System Organ Class, Severity, and Impairment Group

[Implementation Note: A sample figure is shown below. Separate panels will be displayed for each impairment group and matched controls and labeled "Mild Hepatic Impairment (N=X)", "Moderate Hepatic Impairment (N=X)", "Severe Hepatic Impairment (N=X)" and "Matched Controls (N=X)" The y-axis will be labeled "System Organ Class" and the x-axis will be labeled "Number of Events"]



Figure 4: Incidence of Related Adverse Events by MedDRA® System Organ Class, Maximum Severity, and Impairment Group

[Implementation Note: A sample figure is shown below. Separate panels will be displayed for each impairment group and matched controls and labeled "Mild Hepatic Impairment (N=X)", "Moderate Hepatic Impairment (N=X)", "Severe Hepatic Impairment (N=X)" and "Matched Controls (N=X)" The y-axis will be labeled "System Organ Class" and the x-axis will be labeled "Percent of Subjects (%)"]



#### 14.3.5 Displays of Laboratory Results

Figure 5: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – Total Bilirubin



Figures with similar format:

- Figure 6: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group Serum Albumin
- Figure 7 Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group Potassium
- Figure 8: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group Magnesium
- Figure 9: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group Calcium

Figure 10: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Serum Creatinine



Figure 11: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – BUN



Figure 12: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Alkaline Phosphatase



Figure with Similar format:

Figure 13: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – ALT

Figure 14: Chemistry Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Impairment Group – AST


Figure 15: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Hematocrit



#### **Figures with Similar Format:**

Figure 16: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Hemoglobin

Figure 17: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Sex and Impairment Group – Red Blood Cell Count

Figure 18: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – White Blood Cell Count



Figures with Similar Format:

- Figure 19: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group Neutrophils
- Figure 20: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group Eosinophils
- Figure 21: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group Basophils
- Figure 22: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group Lymphocytes
- Figure 23: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group Monocytes
- Figure 24: Hematology Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group Platelets

Figure 25: Coagulation Laboratory Results by Scheduled Visits: Mean Changes from Baseline by and Impairment Group – INR

#### 14.6 Pharmacokinetics

Figure 26: Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Mild Hepatic Impairment



Note: Values below the lower limit of quantification (LLOQ) are plotted as LLOQ/2.

Figures with Similar Format:

Figure 27 Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Moderate Hepatic Impairment

Figure 28: Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Severe Hepatic Impairment

Figure 29: Linear Plot of Pretomanid Concentration Profiles by Nominal Time – Matched Controls

Figure 30: Linear Plot of Pretomanid Concentration Profiles by Nominal Time for Subjects with Mild Hepatic Impairment and Their Matched Controls



Figures with Similar Format:

Figure 31: Linear Plot of Pretomanid Concentration Profiles by Nominal Time for Subjects with Moderate Hepatic Impairment and Their Matched Controls

Figure 32: Linear Plot of Pretomanid Concentration Profiles by Nominal Time for Subjects with Severe Hepatic Impairment and Their Matched Controls

Figure 33: Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time – Mild Hepatic Impairment



Figures with Similar Format:

- Figure 34: Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time Moderate Hepatic Impairment
- Figure 35: Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time Severe Hepatic Impairment
- **Figure 36**: Semilogarithmic Plot of Pretomanid Concentration Profiles by Nominal Time Matched Controls

Figure 37: Linear Plots of Mean Pretomanid Plasma Concentration by Nominal Time



Figure 38: Semilogarithmic Plots of Mean Pretomanid Plasma Concentration by Nominal Time



Figure 39: Impairment Group Summary for Noncompartmental PK Parameters – C<sub>max</sub>

[Implementation Note: Each boxplot may include panels by site if appropriate as described in Section 10.3]



Figure 40: Impairment Group Summary for Noncompartmental PK Parameters – T<sub>max</sub>
 Figure 41: Impairment Group Summary for Noncompartmental PK Parameters – AUC<sub>(0-∞)</sub>
 Figure 42: Impairment Group Summary for Noncompartmental PK Parameters –AUC<sub>(0-last)</sub>
 Figure 43: Impairment Group Summary for Noncompartmental PK Parameters – CL/F
 Figure 44: Impairment Group Summary for Noncompartmental PK Parameters – V<sub>d</sub>/F

## APPENDIX 3. LISTINGS MOCK-UPS

#### **LISTINGS**

| Listing 1: | 16.2.1 Early Terminations or Discontinued Subjects | .184 |
|---|---|---|
| Listing 2: | 16.2.2.1: Subject-Specific Protocol Deviations | .185 |
| Listing 3: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | .186 |
| Listing 4: | 16.2.3: Subjects Excluded from Analysis Populations | .187 |
| Listing 5: | 16.2.4.1: Demographic Data | .188 |
| Listing 6: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | .189 |
| Listing 7: | 16.2.7.2: Unsolicited Adverse Events | .191 |
| Listing 8: | 16.2.8.1: Clinical Laboratory Results – Chemistry | .192 |
| Listing 9: | 16.2.8.2: Clinical Laboratory Results – Hematology | .193 |
| Listing 10: | 16.2.8.3: Clinical Laboratory Results – Urinalysis | .194 |
| Listing 11: | 16.2.8.3: Clinical Laboratory Results – Coagulation | .195 |
| Listing 12: | 16.2.9.1: Vital Signs | .196 |
| Listing 13: | 16.2.9.2: Physical Exam Findings | .197 |
| Listing 14: | 16.2.10: Concomitant Medications | .198 |
| Listing 15: | 16.2.11.1: Pregnancy Reports – Maternal Information | .199 |
| Listing 16: | 16.2.11.2: Pregnancy Reports – Gravida and Para | .199 |
| Listing 17: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | .200 |
| Listing 18: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | .200 |
| Listing 19: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | .200 |
| Listing 20: | Listing of 12-Lead Standard ECG Overall Interpretation and Comments | .201 |
| Listing 21: | Listing of 12-Lead Standard ECG Interval Measurements | .202 |
| Listing 22. | Subject Level Drug Concentrations | 203 |

#### 16.1.6 Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

#### 16.2 Database Listings by Subject

#### **16.2.1 Discontinued Subjects**

#### **Listing 1:** 16.2.1 Early Terminations or Discontinued Subjects

| Impairment Group | Subject ID | Category | Reason for Early Termination | Study Day |
|---|---|---|---|---|

#### **16.2.2 Protocol Deviations**

## **Listing 2:** 16.2.2.1: Subject-Specific Protocol Deviations

| Impairment<br>Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Reason for | Resulted | • | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

**Listing 3:** 16.2.2.2: Non-Subject-Specific Protocol Deviations

| Site | Start Date | Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | <br>Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|

## 16.2.3 Subjects Excluded from the Efficacy Analysis

Listing 4: 16.2.3: Subjects Excluded from Analysis Populations

| Impairment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

#### 16.2.4 Demographic Data

## Listing 5: 16.2.4.1: Demographic Data

| Impairment<br>Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Height at<br>Screening (cm) | Weight at<br>Screening (kg) |
|---|---|---|---|---|---|---|

# Listing 6: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

•

| Impairment<br>Group | MedDRA<br>Preferred<br>Term | MH Number | Medical History Term | Condition Start Day | Condition End Day |
|---|---|---|---|---|---|

## 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not Applicable.

#### 16.2.6 Individual Efficacy/Immunogenicity Response Data

Not Applicable.

#### 16.2.7 Adverse Events

Listing 7: 16.2.7.2: Unsolicited Adverse Events

| Adverse<br>Event | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term | No. of Days<br>Post Dose<br>(Duration) | Severity | SAE? | Relationship to<br>Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| Impairment Group: , Subject ID: , AE Number: | | | | | | | | | | |
| Comments: | | | , | | | | | | | |
| Impairment ( | Group: , Subject ID | : , AE Number: | | | | | | | | |
| Comments: | Comments: | | | | | | | | | |

Note: For additional details about SAEs, see Table 20.

#### 16.2.8 Individual Laboratory Measurements

**Listing 8:** 16.2.8.1: Clinical Laboratory Results – Chemistry

| Impairment<br>Group | Subject ID | Planned<br>Time Point | Actual<br>Study Day | Sex | Laboratory<br>Parameter (Units) | Result (Severity<br>Grade) | Reference<br>Range Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|

#### **Listing 9:** 16.2.8.2: Clinical Laboratory Results – Hematology

| Impairment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|

#### **Listing 10:** 16.2.8.3: Clinical Laboratory Results – Urinalysis

| Impairment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range High |
|---|---|---|---|---|---|---|---|---|---|

#### **Listing 11: 16.2.8.3: Clinical Laboratory Results – Coagulation**

| Impairment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range High |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.9 Vital Signs and Physical Exam Findings

Listing 12: 16.2.9.1: Vital Signs

| Impairment<br>Group | Subject ID | Planned<br>Time Point | Actual<br>Study Time<br>Point | Temperature (°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate (beats/min) | Weight (kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|

#### Listing 13: 16.2.9.2: Physical Exam Findings

| Impairment<br>Group | Planned Time<br>Point | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|

#### **16.2.10** Concomitant Medications

#### **Listing 14:** 16.2.10: Concomitant Medications

| Impairment<br>Group | Subject ID | CM<br>Number | Medication | Medication End<br>Day | Indication | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

**Listing 15:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Impairment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 16: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

#### **Listing 17:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

#### **Listing 18:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress<br>During<br>Labor and<br>Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### Listing 19: 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|

#### Listing 20: Listing of 12-Lead Standard ECG Overall Interpretation and Comments

| Impairment<br>Group | Subject ID | Planned<br>Time Point | Actual Study<br>Time Point | Interpretation | Abnormal Finding | Comments |
|---|---|---|---|---|---|---|

#### **Listing 21: Listing of 12-Lead Standard ECG Interval Measurements**

| Impairment<br>Group | Subject ID | Planned<br>Time Point | Actual Study<br>Time Point | Parameter (units) | Result (Severity) | Change from Baseline |
|---|---|---|---|---|---|---|

#### **Listing 22:** Subject Level Drug Concentrations

| Impairment<br>Group | Subject ID | Nominal Time <sup>a</sup> (hr) | Actual Time <sup>a</sup> (hr) | Drug Concentration (ng/mL) | Sample Within<br>Time Window | Used in λ <sub>z</sub> Calculations | Excluded from NCA | Reason for<br>Exclusion from<br>NCA |
|---|---|---|---|---|---|---|---|---|
| | | | | | yes/no | | | |

<sup>&</sup>lt;sup>a</sup> Times are relative to time of first dose. For actual time, out of window times are indicated by an asterisk.